## 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# Statistical Analysis Plan (Methods)

Protocol Number: VX15-809-115 (Final Analysis - Part A)

A Phase 3, 2-Part, Open-label Study to Evaluate the Safety and Pharmacokinetics of Lumacaftor/Ivacaftor Combination Therapy in Subjects Aged 2 Through 5 Years With Cystic Fibrosis, Homozygous for the *F508del-CFTR* Mutation.

**Author of SAP:** 

Version: 1.0

Version Date of SAP: 23 September 2016

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, MA 02210-1862, USA

#### **CONFIDENTIAL**

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

# 2 TABLE OF CONTENTS

| 1 | Title Page | |
|----|-------------------------------------------------|--------------|
| 2 | Table of Contents | . 2 |
| 4 | Introduction | 5 |
| 5 | Study Objectives | |
| 3 | 5.1 Primary Objective. | |
| | 5.2 Secondary Objectives | |
| | 5.3 Other Objectives | |
| 6 | Study Endpoints | |
| U | 6.1 Primary Endpoint. | |
| | 6.2 Secondary Endpoints | |
| 7 | Study Design | |
| , | 7.1 Overall Design | |
| | 7.2 Sample Size and Power | |
| | 7.3 Randomization. | |
| | 7.4 Blinding and Unblinding | |
| 8 | | |
| | 8.1 All Subjects Set | |
| | 8.2 Safety Set. | |
| 9 | Statistical Analysis | |
| | 9.1 General Considerations | |
| | 9.2 Background Characteristics | 11 |
| | 9.2.1 Subject Disposition | 11 |
| | 9.2.2 Demographics and Baseline Characteristics | 12 |
| | 9.2.3 Prior and Concomitant Medications | 12 |
| | 9.2.4 Study Drug Exposure | 13 |
| | 9.3 Efficacy Analysis | 13 |
| | 9.4 Safety Analysis | 13 |
| | 9.4.1 Adverse Events | 14 |
| | 9.4.2 Clinical Laboratory | 15 |
| | 9.4.3 Electrocardiogram | 15 |
| | 9.4.4 Vital Signs | |
| | 9.4.5 Pulse Oximetry | |
| | 9.4.6 Ophthalmological Examinations | |
| | 9.4.7 Spirometry | |
| | 9.4.8 Physical Examination | 16 |
| | 9.4.9 Other Safety Analysis | |
| 10 | 0 Summary of Interim and IDMC Analyses | 16 |
| 10 | | <b>16</b> 16 |

| 11 References | 16 |
|---|---|
| 12 List of Appendices | 17 |
| Appendix A: Schedule of Assessments | |
| Appendix B: Imputation Rules for Missing Prior/Concomitant Medication Dates | 21 |
| Appendix C: Imputation Rules for Missing AE dates | 22 |
| Appendix D: Criteria for Potentially Clinically Significant Events | |
| Appendix E: Details of Statistical Methodology | |



#### 4 INTRODUCTION

This statistical analysis plan (SAP) is for the final analysis of study VX15-809-115 Part A only and is based on the

- approved clinical study protocol, dated 01 August 2016, Version 2.0,
- approved eCRF, dated 08 June 2016, Version 2.0.

Study VX15-809-115 is a phase 3, 2-part, open-label study to evaluate the safety and pharmacokinetics of lumacaftor/ivacaftor combination therapy in subjects aged 2 through 5 years with cystic fibrosis, homozygous for the *F508del-CFTR* mutation.

This SAP (Methods) documents the planned final safety analysis and data presentation for Part A of VX15-809-115.

SAS® Version 9.2 Software (SAS Institute, Cary, North Carolina, USA) or higher will be used to generate all statistical outputs (tables, figures, listings and datasets).

The SAP will be finalized and approved before the end of Part A with CRFs locked on individual subject basis for the final analysis of Part A. Any changes made to the SAP Methods after the above end of Part A activity has occurred will be documented in the clinical study report for this study.

The analysis addressing the pharmacokinetic (PK) objective of the study will be described in the Clinical Pharmacology Analysis Plan (CPAP) which will be developed separately by the Clinical Pharmacology department at Vertex Pharmaceuticals Incorporated (Vertex).

#### 5 STUDY OBJECTIVES

# 5.1 Primary Objective

#### Part A

To evaluate the PK of lumacaftor (LUM) and ivacaftor (IVA) and their respective metabolites in subjects aged 2 through 5 years with cystic fibrosis (CF), homozygous for F508del

## Part B

To evaluate the safety of LUM/IVA combination therapy in subjects aged 2 through 5 years with CF, homozygous for *F508del* 

# 5.2 Secondary Objectives

#### Part A

To evaluate the safety of LUM/IVA combination therapy in subjects aged 2 through 5 years with CF, homozygous for *F508del* 

#### Part B

- To evaluate the pharmacodynamics (PD) of LUM/IVA combination therapy in subjects aged 2 through 5 years with CF, homozygous for *F508del*
- To evaluate the off-drug PD response after the Washout Period
- To evaluate the PK of LUM and IVA and their respective metabolites in subjects aged 2 through 5 years with CF, homozygous for *F508del*

# 5.3 Other Objectives

Not Applicable

## 6 STUDY ENDPOINTS

# 6.1 Primary Endpoint

### Part A

PK parameters of LUM and IVA

### Part B

Safety and tolerability assessments based on adverse events (AEs), clinical laboratory values (serum chemistry, hematology, coagulation studies, and urinalysis), standard 12-lead electrocardiograms (ECGs), vital signs, pulse oximetry, ophthalmological examinations, and spirometry

# 6.2 Secondary Endpoints

#### Part A

- PK parameters of the metabolites of LUM and IVA
- Safety and tolerability assessments based on AEs, clinical laboratory values (serum chemistry, hematology, coagulation studies, and urinalysis), ECGs, vital signs, pulse oximetry, and spirometry

#### Part B

- Absolute change from baseline in sweat chloride at Week 24
- Absolute change from baseline in body mass index (BMI) and BMI-for-age z-score at Week 24
- Absolute change from baseline in weight and weight-for-age z-score at Week 24
- Absolute change from baseline in stature and stature-for-age z-score at Week 24
- Time-to-first pulmonary exacerbation through Week 24
- Number of pulmonary exacerbations through Week 24
- Number of CF-related hospitalizations through Week 24

- Absolute change in fecal elastase-1 (FE-1) levels from baseline at Week 24
- Absolute change in serum levels of immunoreactive trypsinogen (IRT) from baseline through Week 24
- Change in microbiology cultures from baseline at Week 24
- Absolute change from baseline in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) at Week 24
- Absolute change in sweat chloride from Week 24 at Week 26
- Acceptability/palatability of LUM/IVA granules at Day 1
- Absolute change from baseline in lung clearance index (LCI)<sub>2.5</sub> at Week 24
- Absolute change from baseline in LCI<sub>5.0</sub> at Week 24
- PK parameters of LUM, IVA, and their respective metabolite

### 7 STUDY DESIGN

# 7.1 Overall Design

This is a Phase 3, 2-part, open-label, multicenter study evaluating the PK, safety, tolerability, and PD of multiple doses of LUM/IVA in subjects 2 through 5 years of age (inclusive) with CF, homozygous for *F508del*. Part A is designed to evaluate the PK of LUM and IVA and their respective metabolites and the safety of LUM/IVA combination therapy. Part B is designed to evaluate the safety and PD of LUM/IVA combination therapy and also to evaluate the PK of LUM and IVA and their respective metabolites.

Subjects who participate in Part A may participate in Part B, if they meet the eligibility criteria.

## Part A

Approximately 12 subjects are planned for enrollment. Assuming a 10% dropout rate, approximately 10 subjects should complete Part A. Approximately half of the subjects should complete the study in each of the following weight groups: <14 kg and ≥14 kg at screening. Part A includes the following:

- Screening Period (Day -28 through Day -1)
- Treatment Period (Day 1 through Day  $15 \pm 2$  days)
- Safety Follow-up Visit ( $10 \pm 3$  days after the last dose of LUM/IVA)

Figure 7-1 depicts the schematic for the Part A study design.

A review of safety, tolerability, and available PK data will be completed by an internal Vertex team after Part A to determine the dose(s) to be evaluated in Part B. Additional subjects or treatment cohorts may be enrolled, if data from the initial, planned, 12 subjects are inadequate to make a determination of the dose(s) to be evaluated in Part B.

In the later sections, all discussions and analyses plans will be limited to Part A only.

Figure 7-1 Schematic of Study Design for Part A



IVA: ivacaftor; LUM: lumacaftor; q12h: every 12 hours

Notes: Approximately half of the subjects should complete the study in each of the following weight groups: <14 kg and ≥14 kg at screening. No dose adjustments will be made across the duration of study treatment. On Day 15, only the morning dose of LUM/IVA will be administered.

#### Part B

Approximately 56 subjects are planned for enrollment. Assuming a 10% dropout rate, approximately 50 subjects should complete Part B; at least 10 subjects must be <3 years of age at screening. Subjects should be ≥3 years of age at screening for enrollment in the optional LCI Substudy at a subset of sites. Additional subjects may be enrolled at the sponsor's discretion to achieve up to 30 subjects in the LCI Substudy.

Part B includes the following:

- Screening Period (Day -28 through Day -1)
- Treatment Period (Day 1 through Week  $24 \pm 5$  days)
- Washout Period (Week 24 to Week 26 ± 4 days)
- Safety Follow-up Visit (Week 26 [2 weeks ± 4 days after the last study dose of LUM/IVA])

Figure 7-2 depicts the schematic for the Part B study design.

Subjects who have completed the required visits in Part B may be eligible to enroll in the Treatment Cohort or Observational Cohort of an Extension Study to evaluate long-term treatment with LUM/IVA; enrollment will be based on the eligibility criteria. The Treatment Cohort will enroll subjects who completed LUM/IVA treatment and the Safety Follow-up Visit in Part B. The Observational Cohort will enroll subjects who received at least 4 weeks of LUM/IVA treatment in Part B and completed visits up to the Safety Follow-up Visit, if applicable, in Part B, but do not meet eligibility criteria for enrollment into the Treatment Cohort. The Safety Follow-up Visit, if applicable, is the last visit for Part B, and should also be the Day 1 Visit in the Extension Study.

Figure 7-2 Schematic of Study Design for Part B



ETT: Early Termination of Treatment; IVA: ivacaftor; LCI: lung clearance index; LUM: lumacaftor; q12h: every 12 hours Notes: Approximately 56 subjects are planned for enrollment. Assuming a 10% dropout rate, approximately 50 subjects should complete Part B; at least 10 subjects must be <3 years of age. Subjects should be ≥3 years of age for enrollment in the optional LCI Substudy at a subset of sites. Additional subjects may be enrolled at the sponsor's discretion to achieve up to 30 subjects in the LCI Substudy.

- The doses listed above are the planned doses for Part B. Depending on the results from Part A, a single dose from Part A may be selected for all subjects in Part B or a previously unspecified dose or doses may be selected for Part B. No dose adjustments across the duration of treatment will be made. The last dose of LUM/IVA in Part B will be the evening dose before the Week 24 Visit.
- Subjects who prematurely discontinue LUM/IVA treatment will be asked to complete the ETT Visit, to remain on study, and to complete the study assessments from the time of LUM/IVA discontinuation through the Week 24 Visit and the Safety Follow-up Visit, if applicable. The Safety Follow-up Visit is not required for subjects who permanently discontinue LUM/IVA treatment before or at the Week 16 Visit if they return for the Week 24 Visit or for subjects who continue onto commercially-available LUM/IVA by prescription of a physician within 2 weeks (± 4 days) of completing LUM/IVA treatment at Week 24 or at the ETT Visit.
- Subjects who have completed the required visits in Part B may be eligible to enroll in the Treatment Cohort or Observational Cohort of an Extension Study to evaluate long-term treatment with LUM/IVA; enrollment will be based on the eligibility criteria.

# 7.2 Sample Size and Power

No formal sample size calculations have been performed for Part A. The number of subjects participating is common in early clinical pharmacology studies and is considered sufficient to achieve the PK objectives of Part A.

#### 7.3 Randomization

Part A is an open-label study with weight-based treatment group assignment. Randomization is not required in this Part.

# 7.4 Blinding and Unblinding

This is an open-label study. However for Part A, subjects and their legally appointed and authorized representative (e.g., parent or legal guardian) should not be informed of their study-related spirometry (subjects  $\geq 3$  years of age at corresponding part's screening) during the study, regardless if the subject permanently discontinues treatment.

## 8 ANALYSIS SETS

# 8.1 All Subjects Set

All Subjects Set is defined as all subjects who have signed informed consent (and assent, if applicable) and enrolled or dosed in Part A. This analysis set will be used for all individual subject data listings and the disposition summary table, unless specified otherwise.

# 8.2 Safety Set

Safety Set will include all subjects who received at least 1 dose of study drug in Part A. The Safety Set will be used for all safety analyses, with subjects analyzed according to the treatment they received, unless specified otherwise. In addition, the summary by the dosing groups (LUM 100 mg/IVA 125 mg q12h and LUM 150 mg/IVA 188 mg q12h) at enrollment determined by weight at the Screening Visit will be provided as supplementary information.

#### 9 STATISTICAL ANALYSIS

# 9.1 General Considerations

The Schedule of Assessments is provided in Appendix A. The precision standards for reporting safety variables are provided in an internal Biometrics document that specifies the programming rules including the precision for derived variables.

All individual subject data based on All Subjects Set of the corresponding part will be presented in data listings.

Continuous variables will be summarized using the following descriptive summary statistics: number of subjects (n), mean, standard deviation (SD), standard error (SE), median, minimum (min), and maximum (max).

Categorical variables will be summarized using counts and percentages.

Baseline value, unless specified otherwise, will be defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug. For

ECGs, the baseline value will be defined as the average of the pretreatment measurements on Day 1.

Change (absolute change) from baseline will be calculated as postbaseline value - baseline value.

**Relative change from baseline**: will be calculated and presented in percentage as  $100 \times (postbaseline \ value - baseline \ value)/baseline \ value$ .

**Treatment-emergent Period for Part A** will include the time period starting from the first dose date of the study drug through 14 days after last dose of study drug. The Treatment-Emergent period will be used for safety analyses unless specified otherwise.

**Unscheduled visits:** Unscheduled visit measurements will be included in analysis as follows:

- In the derivation of baseline measurements.
- In individual subject data listings as appropriate.

**Visit windowing rules:** The majority of assessments are anticipated to be on schedule. Visit windowing will not add significant value to the analysis and will not be applied. Nominal visit will be used for all assessments.

Incomplete/missing data will not be imputed, unless specified otherwise.

**Outliers:** No formal statistical analyses will be performed to detect or remedy the presence of statistical outliers, unless specified otherwise.

**Multiplicity:** No multiplicity adjustment will be performed and there is no hypothesis testing.

Unless otherwise specified, the analysis will be performed using descriptive summary statistics by dosing groups (LUM 100 mg/IVA 125 mg q12h and LUM 150 mg/IVA 188 mg q12h) and overall. All summaries will be based on the Safety Set. No statistical hypothesis testing will be performed.

# 9.2 Background Characteristics

# 9.2.1 Subject Disposition

The number of subjects in the following categories will be summarized by dosing group and overall:

- All Subjects Set
- Dosed (Safety Set)

The numbers and percentages (based on the Safety Set) of subjects in the following disposition categories will be summarized by dosing group and overall

- Completed study drug treatment
- Prematurely discontinued the treatment and the reasons for discontinuations
- Completed study
- Prematurely discontinued the study and the reasons for discontinuations

A listing will be provided for subjects who discontinued treatment or who discontinued study with reasons for discontinuation.

# 9.2.2 Demographics and Baseline Characteristics

Demographics, medical history and baseline characteristics will be summarized overall and by dosing group based on the Safety Set.

Demographic data will include the following:

- Age at baseline
- Sex (female and male)
- Ethnicity (Hispanic or Latino, not Hispanic or Latino, and not collected per local regulations)
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, and Other)

Baseline characteristics will include the following:

- Weight (kg)
- Stature (cm)
- BMI (kg/m2)

Medical history will be summarized by MedDRA system organ class (SOC) and preferred term (PT).

## 9.2.3 Prior and Concomitant Medications

Medications used in this study will be coded by using the World Health Organization Drug Dictionary Enhanced (WHODDE) and categorized as the following:

- **Prior medication:** any medication that started before initial dosing of study drug in each part, regardless of when it ended.
- Concomitant medication: medication continued or newly received at or after initial dosing of study drug in each part to 14 days after the last dose of study drug in the corresponding part.
- **Post-treatment medication:** medication continued or newly received after 14 days after the last dose of study drug in each part.

A given medication can be classified as a prior medication, a concomitant medication, or a post-treatment medication; both prior and concomitant; both concomitant and post-treatment; or prior, concomitant, and post-treatment.

If a medication has a missing or partially missing start/end date or time and it cannot be determined whether it was taken before initial dosing, concomitantly, or after 14 days after the last dose of study drug, it will be considered as prior, concomitant, and post-treatment.

Prior medications and concomitant medications will be summarized descriptively by 1) preferred names; 2) anatomic class (ATC) level 1, ATC level 2, and preferred names based on the Safety Set.

Summaries of medications will be based on the Safety Set.

Details for imputing missing or partial start and/or stop dates of medication are described in Appendix B.

# 9.2.4 Study Drug Exposure

Duration of study drug exposure is defined as follows: last dose date – first dose date + 1 day, regardless of any interruptions in dosing. If the last dose date of study drug is missing, the subject's last date from the dosing panel (excluding PK dosing) will be used for analysis purposes.

Study drug exposure will be summarized descriptively (n, mean, SD, SE, median, min, and max in days) by dosing group and overall based on Safety Set. In addition, the summary by the dosing group (LUM 100 mg/IVA 125 mg q12h and LUM 150 mg/IVA 188 mg q12h) at enrollment determined by weight at the Screening Visit will be provided as supplementary information.

Study drug exposure will be presented in an individual subject data listing to indicate whether the study drug was taken or not.

# 9.3 Efficacy Analysis

Not Applicable

# 9.4 Safety Analysis

The overall safety profile of study drug will be assessed in terms of the following safety and tolerability endpoints:

- Incidence of treatment-emergent adverse events (TEAEs)
- Clinical laboratory values (serum chemistry, hematology, coagulation studies, and urinalysis)
- ECGs (standard 12-lead)
- Vital signs
- Pulse oximetry
- Spirometry (subjects  $\geq 3$  years age at screening)

Safety analyses will be performed by dosing group and overall. Safety analyses will be conducted for the Safety Set. Safety data will be presented in the individual subject data listings based on the All Subjects Set. Only descriptive summary statistics of safety data will be provided (i.e., no statistical hypothesis testing will be performed).

The summary by the dosing groups (LUM 100 mg/IVA 125 mg q12h and LUM 150 mg/IVA 188 mg q12h) at each part's enrollment determined by weight at the Screening Visit will be provided as the supplementary information.

## 9.4.1 Adverse Events

AEs will be classified as pretreatment AEs, TEAEs, or post-treatment AEs.

- Pretreatment AE: any AE that started before initial dosing of study drug in each part.
- **TEAE**: any AE that increased in severity or that was newly developed during the Treatment Period which is defined as being the period from initial dosing of study drug in each part to 14 days after the last dose of study drug in the corresponding part.
- **Post-treatment AE**: any AE that increased in severity or that developed after 14 days after the last dose of study drug in each part.

For AEs with missing or partial start dates, if there is no clear evidence that the AEs started before or after study treatment, then the AEs will be classified as TEAEs.

Details for imputing missing or partial start dates of adverse events are described in Appendix C.

TEAE summaries will be presented using number and percentages of subjects.

An overview of TEAE profile will be provided, including total number of TEAEs, with number and percentage of subjects for the following categories: (1) All TEAEs, (2) Grades 3/4 TEAEs, (3) TEAEs by relationship to study drug, (4) TEAEs by maximum severity, (5) TEAEs leading to treatment interruption, (6) TEAEs leading to treatment discontinuation, (7) Serious TEAEs, (8) Serious TEAEs related to study drug, and (9) TEAEs leading to death.

AE summary tables will be presented for TEAEs only and will include the following:

- All TEAEs
- Grades 3/4 TEAEs
- TEAEs by relationship to study drug
- TEAEs by maximum severity
- TEAEs leading to treatment interruption
- TEAEs leading to treatment discontinuation
- Serious TEAEs
- Serious TEAEs related to study drug
- TEAEs leading to death

Summaries will be presented by MedDRA system organ class (SOC) and preferred term (PT) using frequency counts and percentages. When summarizing the number and percentage of subjects with an event, subjects with multiple occurrences of the same AE or a continuing AE will be counted once, only the maximum severity level will be presented in the severity summaries, and the worst/highest relationship level in the relationship summaries.

Separate tables will be provided summarizing the number of subjects, the number of events and the number of related events for the following by SOC and PT as per EudraCT requirement:

- Treatment-emergent Serious AEs
- Treatment-emergent Non-Serious AEs

Note if an event increases in its severity, it will be reported as a separate event in the clinical database and thus may be counted more than once.

In addition, listings that contain individual subject data for all TEAEs leading to treatment interruption, TEAEs leading to treatment discontinuation, deaths, and serious AEs will be provided separately. All AEs, including pre- and post-treatment AEs, will be presented in individual subject data listings.

# 9.4.2 Clinical Laboratory

For laboratory measurements, the raw values and change from baseline values of the continuous hematology/coagulation and chemistry results will be summarized by dosing group and overall in SI units at each scheduled time point. For hematology and chemistry, the number and percentage of subjects with abnormal low (<lower limit of normal [LLN]) value and with abnormal high (>ULN) value at each scheduled time point will be summarized.

The number and percentage of subjects with at least 1 potentially clinically significant (PCS) laboratory event (i.e., categorical change) during the Treatment-Emergent period will be summarized. The PCS/categorical criteria are provided in Appendix D.

Results of urinalysis will be listed in individual subject data listings only.

In addition, a listing containing individual subject hematology, chemistry, and coagulation values outside the normal reference ranges will be provided. This listing will include data from both scheduled and unscheduled visits.

## 9.4.3 Electrocardiogram

For ECG measurements, a summary of raw values and change from baseline values will be provided by dosing group and overall at each scheduled time point for the following standard 12-lead ECG measurements: RR (ms), HR (bpm), PR (ms), QRS duration (ms), QT (ms), and QT corrected for HR intervals [Fridericia's correction QTcF (ms) =QT/RR<sup>1/3</sup>]. In addition, the mean value at each time point will be plotted for QTcF.

The number and percentage of subjects with at least 1 PCS ECG event (i.e., categorical change) during the Treatment-Emergent period will be summarized. The PCS/categorical criteria are provided in Appendix D.

The number and percentage of subjects with shift changes from baseline (normal/missing, not clinically significant, and potentially clinically significant according to overall ECG evaluation) to the worst ECG evaluation during the Treatment Period will be summarized.

# 9.4.4 Vital Signs

For vital signs measurements, the raw values and change from baseline values will be summarized by dosing group and overall at each scheduled time point: systolic and diastolic blood pressure (mm Hg), body temperature (°C), pulse rate (beats per minute), and respiratory rate (breaths per minute).

The number and percentage of subjects with at least 1 PCS vital sign event (i.e., categorical change) during the Treatment period will be summarized. The PCS/categorical criteria are provided in Appendix D.

# 9.4.5 Pulse Oximetry

For the pulse oximetry measurements, a summary of raw values and change from baseline values will be provided at each scheduled time point for the percent of oxygen saturation by pulse oximetry.

The number and percentage of subjects with shift changes from baseline (normal/missing and low according to the reference range) to the lowest percent of oxygen saturation during the Treatment Period will be provided.

# 9.4.6 Ophthalmological Examinations

Ophthalmological examination findings (Screening only) will be presented as a data listing.

# 9.4.7 Spirometry

Spirometry data will be presented as a data listing only.

# 9.4.8 Physical Examination

Physical examination findings will be presented as a data listing only.

# 9.4.9 Other Safety Analysis

Not applicable.

#### 10 SUMMARY OF INTERIM AND IDMC ANALYSES

# 10.1 Interim Analysis

No interim analysis is planned but interim analyses may take place at any time during the study if warranted by the ongoing data, and/or deemed necessary by the internal Vertex team.

## 10.2 IDMC Analysis

Details of the IDMC (Section 8.2 of the protocol) analysis will be provided in the IDMC Analysis Plan. There is no IDMC analysis for Part A.

## 11 REFERENCES

<sup>1</sup>Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall G, Culver BH, et al. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012;40(6):1324-43.

# 12 LIST OF APPENDICES

**Appendix A: Schedule of Assessments** 

Table 12-1 Study VX15-809-115: Part A Screening

| Assessment | Screening Visit Day -28 through Day -1 |
|---|---|
| Informed consent/assent | X |
| Demographics | X |
| Medical and ophthalmological history | X |
| Stature, weight, and vital signs <sup>a,b</sup> | X |
| Pulse oximetry <sup>b</sup> | X |
| Ophthalmologic examination <sup>c</sup> | X |
| Full physical examination | X |
| Standard 12-lead ECG <sup>d</sup> | X |
| Spirometry <sup>e</sup> | X |
| CFTR genotype <sup>f</sup> | X |
| Serum chemistry <sup>g</sup> | X |
| Hematology <sup>g</sup> | X |
| Coagulation studies <sup>g</sup> | X |
| Urinalysis <sup>g</sup> | X |
| Medications review <sup>h</sup> | Continuous from signing of ICF through Safety Follow-up Visit |
| Adverse events | Continuous from signing of ICF through Safety Follow-up Visit |

BMI: body mass index; CFTR: cystic fibrosis transmembrane conductance regulator gene; ECG: electrocardiogram; ICF: informed consent form.

<sup>a</sup> If children can stand unassisted and follow directions, stature should be measured as height; otherwise, stature will be measured as length. Stature and weight must be measured with shoes off and while wearing light clothing. BMI will be derived from this assessment. Refer to Section 11.4.3 of the protocol for details.

The subject should rest for at least 5 minutes before having vital signs and pulse oximetry measured. Refer to Section 11.6.4 of the protocol for details.

An ophthalmologic examination will be conducted by a licensed ophthalmologist. The examination does not need to be repeated if there is documentation of an examination meeting protocol criteria that was conducted within 3 months before the Screening Visit. Subjects with documentation of bilateral lens removal do not need the ophthalmologic examination. Refer to Section 11.6.6 of the protocol for details.

A standard 12-lead ECG will be performed. The subject will be instructed to rest in the supine position for at least 5 minutes, if possible, before having an ECG performed. The ECG will be performed before any other procedures that may affect heart rate, such as blood draws. Refer to Section 11.6.5 of the protocol for details.

<sup>e</sup> Spirometry (subjects ≥3 years of age at screening only) may be performed pre- or post-bronchodilator. Refer to Section 11.6.7 of the protocol for details.

All subjects will be tested to assess *CFTR* genotype, regardless of availability of a previous *CFTR* genotype laboratory report. Refer to Section 11.6.2 of the protocol for details.

Refer to Section 11.6.2 of the protocol for details.

h Refer to Section 9.4.2 of the protocol for details.

Study VX15-809-115: Part A Treatment Period and Safety Follow-up Visit **Table 12-2** 

| | | Day 3 | Day 8 | Day 15 | Safety Follow-up Visit<br>10 (± 3) Days After the Last |
|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Day 1 | (± 1 Day) | $(\pm 1 \text{ Day})$ | $(\pm 2 \text{ Days})$ | Dose of Study Drug |
| Clinic visit | X | | X | X | X |
| Telephone contact <sup>b</sup> | | X | | | |
| Safety Assessments | | | | | |
| Stature and weight <sup>c</sup> | X | | | X | X |
| Vital signs <sup>d</sup> | X | | X | X | X |
| Pulse oximetry <sup>d</sup> | X | | X | X | X |
| Full physical examination <sup>e</sup> | X | | | X | X |
| Standard 12-lead ECG <sup>f</sup> | $X^g$ | | | Xg | X |
| Spirometry <sup>h</sup> | X | | X | X | X |
| Serum chemistry <sup>i</sup> | X | | X <sup>i</sup> (LFT only) | X | X |
| Hematology <sup>j</sup> | X | | | X | X |
| Coagulation studies <sup>i</sup> | X | | | X | X |
| Urinalysis <sup>i</sup> | X | | | X | X |
| | | | | | NAME AND ADDRESS OF THE PARTY O |

All assessments will be performed before LUM/TVA dosing unless noted otherwise (Section 11.1 of the protocol). When repeats of an assessment are required postdose at a given visit, the assessment will be collected only once if LUM/IVA is not administered on the day of the visit (i.e., LUM/IVA interruption or permanent LUM/IVA

Liver function testing (ALT, AST, GGT, ALP, and total bilirubin) will be performed at the Day 8 Visit. Refer to Section 11.6.2 of the protocol for details.

Refer to Section 11.6.2 of the protocol for details.

Telephone contact will be made to assess the subject's status, any AEs, concomitant medications, treatments, and procedures.

If children can stand unassisted and follow directions, stature should be measured as height; otherwise, stature will be measured as length. Stature and weight must be measured with shoes off and while wearing light clothing. BMI will be derived from this assessment. Refer to Section 11.4.3 of the protocol for details.

Symptom-directed physical examinations will occur at any time during the study if triggered by AEs or if deemed necessary by the investigator. Refer to Section 11.6.4 The subject should rest for at least 5 minutes before having vital signs and pulse oximetry measured. Refer to Section 11.6.4 of the protocol for details.

performed. The ECG will be performed before any other procedures that may affect heart rate, such as blood draws. Refer to Section 11.6.5 of the protocol for details. A standard 12-lead ECG will be performed. The subject will be instructed to rest in the supine position for at least 5 minutes, if possible, before having an ECG of the protocol for details.

Standard 12-lead ECGs will be performed at the following times: at the Day 1 and Day 15 Visits before the morning dose of LUM/IVA, and at 1.5, 3, 4, and 6 hours after Spirometry (subjects  $\geq$ 3 years of age at screening only) should be performed pre-bronchodilator. On Day 1, spirometry will be performed before the morning dose and the morning dose of LUM/IVA. Predose ECGs on Day 1 will be performed in triplicate. A window of ± 15 minutes will be allowed around the nominal times for all postdose ECG assessments.

<sup>4</sup> hours (±30 minutes) after the morning dose of LUM/IVA. On Day 8 and Day 15, spirometry will be performed before the morning dose of LUM/IVA. Refer to Section 11.6.7 of the protocol for details.

Vertex Pharmaceuticals Incorporated

Study VX15-809-115: Part A Treatment Period and Safety Follow-up Visit **Table 12-2** 

| | | Day 3 | Day 8 | Day 15 | Safety Follow-up Visit 10 ( $\pm$ 3) Days After the Last |
|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Day 1 | (± 1 Day) | (± 1 Day) | $(\pm 2 \text{ Days})$ | Dose of Study Drug |
| Observation 4 hours after the first dose | X | | | | |
| Medications, treatments, and procedures reviewk | Continuous from | I do guingis of I | Continuous from signing of ICF through Safety Follow-up Visit | 'ollow-up Visit | |
| Adverse events | Continuous from | I do guingis I | Continuous from signing of ICF through Safety Follow-up Visit | 'ollow-up Visit | |
| PK Assessments | | | | | |
| PK sampling | $X^{l}$ | | $X_{\mathrm{m}}$ | $_{ m u} { m X}$ | |
| Study Drug Administration | | | | | |
| | | IT | LUM/IVA q12h | | |
| LUM/IVA dosing° | Day 1 thr | ough Day 1: | Day 1 through Day 15 (morning dose only on Day 15) | ly on Day 15) | |
| AF: adverse event: ALP: alkaline phosphatase: ALT: alanine aminotransferase: AST: aspartate aminotransferase: BMI: body mass index: CF: cyclic fibrosis: | ninotransferase: | AST: aspa | rtate aminotransfers | se: BMI: body n | nass index: CF: evstie fibrosis: |

AE: adverse event, ALE: atkaline phosphatase; AL1: atanine animotransferase; AS1: aspartate animotransferase; DMI: body mass moex; CF: cystic norosis; ECG: electrocardiogram; GGT: gamma glutamyl transpeptidase; ICF: informed consent form; IVA: ivacaflor; LFT: liver function testing; LUM: lumacaflor; PK: pharmacokinetic; q12h: every 12 hours

Refer to Section 9.4.2 of the protocol for details.

On Day 1, a PK blood sample will be collected at 3 to 4 hours after the morning dose of LUM/IVA. Refer to Section 11.3.1 of the protocol for details.

On Day 8, PK blood samples will be collected predose (within 60 minutes before the morning dose). Refer to Section 11.3.1 of the protocol for details.

On Day 15, a PK blood samples will be collected predose (within 60 minutes before the morning dose), and 2 hours (± 15 minutes) and 3 to 4 hours after the morning dose of LUM/IVA. Refer to Section 11.3.1 of the protocol for details.

LUM/IVA will be administered q12h (± 1 hour), approximately 30 minutes from the start of consuming fat containing food such as a standard "CF" high fat, high calorie meal or snack according to the guidelines in Section 10.2.1 of the protocol. The morning dose on Day 15 is the last dose of LUM/IVA.

# **Appendix B: Imputation Rules for Missing Prior/Concomitant Medication Dates**

Imputation rules for missing or partial medication start/stop dates are defined below:

- 1. Missing or partial medication start date:
  - a. If only DAY is missing, use the first day of the month.
  - b. If DAY and Month are both missing, use the first day of the year.
  - c. If DAY, Month and Year are all missing, use a date before the first dose date.
- 2. Missing or partial medication stop date:
  - a. If only DAY is missing, use the last day of the month.
  - b. If DAY and Month are both missing, use the last day of the year.
  - c. If DAY, Month and year are all missing, assign 'continuing' status to stop date.

In summary, the prior, concomitant or post categorization of a medication is described below.

Table 12-3 Prior, Concomitant, and Post Categorization of a Medication

| | | <b>Medication Stop Date</b> | |
|---|---|---|---|
| Medication Start Date | < First Dose Date of<br>Study Drug | ≥ First Dose Date<br>and ≤ End Date of<br>Treatment-emergent<br>Period | > End Date of<br>Treatment-emergent<br>Period |
| < First dose date of study drug | P | PC | PCA |
| ≥ First dose date and<br>≤ End date of Treatment-<br>emergent period | - | С | CA |
| > End date of Treatment-<br>emergent period | - | - | A |

A: Post; C: Concomitant; P: Prior

# Appendix C: Imputation Rules for Missing AE dates

Imputation rules for missing or partial AE start date are defined below:

# If only Day of AE start date is missing:

If the AE start year and month are the same as that for the first dose date, then:

- If the full (or partial) AE end date is NOT before the first dose date or AE end date is missing, then impute the AE start day as the day of first dose date; otherwise, impute the AE start day as 1.
- Otherwise, impute the AE start day as 1.

Compare the imputed AE start date with Treatment-Emergent period to determine whether the AE is pretreatment AE, TEAE or post-treatment AE.

# If Day and Month of AE start date are missing:

If AE start year = first dose year, then:

- If the full (or partial) AE end date is NOT before the first dose date or AE end date is missing, then impute the AE start Month and Day as the Month and Day of first dose date; otherwise, impute the AE start Month as January and the Day as 1.
- Otherwise, impute the AE start MONTH as January and the DAY as 1.

Compare the imputed AE start date with Treatment-Emergent period to determine whether the AE is pretreatment AE, TEAE or post-treatment AE.

# If Year of AE start date is missing:

If the year of AE start is missing or AE start date is completely missing then query site with no imputation. Also compare the full (or partial) AE end date to the first dose date. If the AE end date is before the first dose date then the AE should be considered as a pretreatment AE. Otherwise, the AE will be considered as TEAE.

# **Appendix D: Criteria for Potentially Clinically Significant Events**

 Table 12-4
 Criteria for Potentially Clinically Significant Laboratory Tests

| Parameter | PCS | Comments |
|---|---|---|
| Clinical Chemistr | y | |
| ALT | ≤3xULN*(Not a PCS criterion) >3x - ≤ 5xULN >5x - ≤ 8xULN >3xULN >5xULN >8xULN | FDA DILI Guidance Jul 2009. |
| AST | ≤3xULN*(Not a PCS criterion) >3x - ≤ 5xULN >5x - ≤ 8xULN >3xULN >5xULN >8xULN | FDA DILI Guidance Jul 2009. |
| ALT or AST | ALT>3xULN or AST>3xULN | Vertex LFT working group 2014 |
| Alkaline<br>Phosphatase | >1.5xULN | FDA DILI Guidance Jul 2009. |
| Total Bilirubin | >1.5x - ≤2xULN<br>>2xULN | FDA DILI Guidance Jul 2009. |
| ALT and Total<br>Bilirubin | ALT>3xULN and TBILI>2xULN | FDA DILI Guidance Jul 2009. To be counted within a same treatment phase, whatever the interval between measurements. |
| AST and Total<br>Bilirubin | AST>3xULN and TBILI>2xULN | FDA DILI Guidance Jul 2009. To be counted within a same treatment phase, whatever the interval between measurements. |
| (ALT or AST) and<br>Total Bilirubin | (ALT>3xULN or AST>3xULN) and TBILI>2×ULN | Vertex LFT working group 2014 |
| СРК | >3x - ≤ 10xULN<br>>10xULN | FDA criteria Feb 2005.<br>Am J Cardiol April 2006. |
| Creatinine | ≥150 µmol/L (Adults)<br>≥30% change from baseline<br>≥100% change from baseline | Benichou C., 1994. |
| Blood Urea<br>Nitrogen | ≥17 mmol/L | |
| Chloride | <85 mmol/L<br>>115 mmol/L | |
| Sodium | $\leq$ 129 mmol/L $\geq$ 150 mmol/L | |
| Potassium | <3 mmol/L<br>≥5.5 mmol/L | FDA Feb 2005. |

Table 12-4 Criteria for Potentially Clinically Significant Laboratory Tests

| Parameter | PCS | Comments |
|---|---|---|
| Glucose | | |
| Hypoglycaemia | ≤3.9 mmol/L and <lln< td=""><td>ADA May 2005.</td></lln<> | ADA May 2005. |
| Hyperglycaemia | $\geq$ 11.1 mmol/L (unfasted); $\geq$ 7 mmol/L (fasted) | ADA Jan 2008. |
| Albumin | ≤25 g/L | |
| Hematology | | |
| WBC | <3.0 Giga/L (Non-Black); <2.0 Giga/L (Black) ≥16.0 Giga/L | Increase in WBC: not relevant. To be interpreted only if no differential count available. |
| Lymphocytes | >4.0 Giga/L | |
| Neutrophils | <1.5 Giga/L (Non-Black);<1.0 Giga/L (Black) | International Consensus meeting on drug-<br>induced blood cytopenias, 1991.<br>FDA criteria. |
| Monocytes | >0.7 Giga/L | |
| Basophils | >0.1 Giga/L | |
| Eosinophils | >0.5 Giga/L or >ULN (if ULN≥0.5 Giga/L) | Harrison- Principles of internal Medicine 17th Ed., 2008. |
| Hemoglobin | ≤115 g/L (Male); ≤95 g/L (Female)<br>≥185 g/L (Male); ≥165 g/L (Female)<br>Decrease from Baseline ≥20 g/L | Criteria based upon decrease from baseline are more relevant than based on absolute value. Other categories for decrease from baseline can be used (≥30 g/L, ≥40 g/L, |
| | Decreuse from Busenine -20 g/E | ≥50 g/L). |
| Hematocrit | ≤0.37 v/v (Male) ; ≤0.32 v/v (Female)<br>≥0.55 v/v (Male) ; ≥0.5 v/v (Female) | |
| RBC | ≥6 Tera/L | |
| Platelets | <100 Giga/L<br>≥700 Giga/L | International Consensus meeting on drug-<br>induced blood cytopenias, 1991. |

Table 12-5 Criteria for Potentially Clinically Significant ECGs

| Parameter | PCS | Comments |
|---|---|---|
| HR | ≤50 bpm and decrease from baseline ≥20 bpm<br>≥120 bpm and increase from baseline ≥20 bpm | |
| PR | ≥220 ms and increase from baseline ≥20 ms | 1 |
| QRS | ≥120 ms | |

Table 12-5 Criteria for Potentially Clinically Significant ECGs

| Parameter | PCS | Comments |
|---|---|---|
| QTc | Absolute values (ms) | To be applied to any kind of QT correction |
| Borderline | Borderline: 431-450 ms (Male); 451-470 ms | formula. |
| Prolonged* | (Female) | |
| Additional | Prolonged: >450 ms (Male); >470 ms (Female) | |
| | ≥500 ms | |
| | Increase from baseline | |
| | Borderline: Increase from baseline 30-60 ms | |
| | Prolonged: Increase from baseline >60 ms | |

Note: Based on CPMP 1997 guideline.

Table 12-6 Criteria for Potentially Clinically Significant Vital Signs

| Parameter | PCS | Comments |
|---|---|---|
| HR | ≤50 bpm and decrease from baseline ≥20 bpm ≥120 bpm and increase from baseline≥20 bpm | To be applied for all positions (including missing) except STANDING. |
| SBP | ≤95 mmHg and decrease from baseline<br>≥20mmHg<br>≥160 mmHg and increase from baseline ≥20<br>mmHg | To be applied for all positions (including missing) except STANDING. |
| DBP | ≤45 mmHg and decrease from baseline ≥10 mmHg ≥110 mmHg and increase from baseline ≥10 mmHg | To be applied for all positions (including missing) except STANDING. |
| Weight | ≥5% increase from baseline<br>≥5% decrease from baseline | FDA criteria Feb 2007. |

# Appendix E: Details of Statistical Methodology

Percent predicted values will be calculated for parameters of FEV<sub>1</sub>, FVC, FEV1/FVC, and FEF<sub>25%-75%</sub> using the Quanjer GLI-2012 Regression Equations and Lookup Tables.

The regression equations and lookup tables required to implement the Quanjer GLI-2012 predicted values are available in:

Quanjer GLI-2012 Regression Equations and Lookup Tables. Philip H. Quanjer, Sanja Stanojevic, Tim J. Cole, Janet Stocks. Version 7 April 2013. Available at: http://www.erseducation.org/guidelines/global-lung-function-initiative/tools/quanjer-gli-2012-regression-equations-and-lookup-tables.aspx. Accessed 08 December 2015.

The instructions and tools on how to implement the Quanjer GLI-2012 equations are:

Implementing GLI-2012 regression equations. Philip H. Quanjer, Sanja Stanojevic, Tim J. Cole, Janet Stocks. Version 19 July 2015. Available at: http://www.erseducation.org/guidelines/global-lung-function-initiative/gli-2012-explained.aspx. Accessed 08 December 2015.

GLI-2012 - SAS Macro. Sanja Stanojevic. Version 2, 7 April 2013. Available at: http://www.ers-education.org/guidelines/global-lung-function-initiative/tools/sas-macro.aspx. Accessed 08 December 2015.

## 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# Statistical Analysis Plan (Methods)

Protocol Number: VX15-809-115 (Final Analysis - Part B)

A Phase 3, 2-Part, Open-label Study to Evaluate the Safety and Pharmacokinetics of Lumacaftor/Ivacaftor Combination Therapy in Subjects Aged 2 Through 5 Years With Cystic Fibrosis, Homozygous for the *F508del-CFTR* Mutation.

**Author of SAP:** 



Version: 2.0 Version Date of SAP: 07 September 2017

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, MA 02210-1862, USA

#### **CONFIDENTIAL**

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

## 2 TABLE OF CONTENTS

Table of Contents

1

| | 1 661 | Die di Contenty | |
|---|-------|-----------------------------------------------|----|
| 4 | Int | roduction | 5 |
| 5 | Stu | ıdy Objectives | 5 |
| | 5.1 | Primary Objective | 5 |
| | 5.2 | Secondary Objectives | 5 |
| | 5.3 | Other Objectives | 6 |
| 6 | Stu | idy Endpoints | 6 |
| | 6.1 | Primary Endpoint. | 6 |
| | 6.2 | J = -1 | |
| 7 | | ıdy Design | |
| | 7.1 | Overall Design | |
| | 7.2 | Randomization | |
| | 7.3 | Blinding and Unblinding | |
| 8 | | alysis Sets | |
| | 8.1 | All Subjects Set | |
| | 8.2 | Safety Set | |
| | 8.3 | Full Analysis Set. | |
| | 8.4 | LCI Substudy Set. | |
| 9 | Sta | tistical Analysis | |
| | 9.1 | General Considerations | |
| | 9.2 | Background Characteristics | |
| | 9.2 | 2.1 Subject Disposition | |
| | 9.2 | 2.2 Demographics and Baseline Characteristics | 13 |

Prior and Concomitant Medications 14

Adverse Events 16

Electrocardiogram 19

Ophthalmological Examinations 20

Other Safety Analysis 21

923

9.2.4

9.2.5

926

9.4.1

9.4.2

9.4.3

9.4.4

9.4.5

9.4.6

9.4.7

9.4.89.4.9

9.3

9.4

| | 9.5 Pharma | codynamic Analysis | 21 |
|---|---|---|---|
| | | nalysis of Primary Endpoints | |
| | | nalysis of Secondary Pharmacodynamic Endpoints | |
| | 9.5.2.1 | Absolute Change From Baseline in Sweat Chloride at Week 24 | |
| | 9.5.2.2 | Absolute Change From Baseline in BMI/BMI-for-Age Z-score at | |
| | | Week 24 | 22 |
| | 9.5.2.3 | Absolute Change From Baseline in Weight/Weight-for-Age Z-Score at | |
| | | Week 24 | 22 |
| | 9.5.2.4 | Absolute Change From Baseline in Stature/Stature-for-Age Z-score at | |
| | | Week 24 | 23 |
| | 9.5.2.5 | Analysis of Pulmonary Exacerbation-related Other Secondary | |
| | | Pharmacodynamic Variables. | |
| | 9.5.2.6 | Absolute Change in FE-1 Levels From Baseline at Week 24 | 23 |
| | 9.5.2.7 | Absolute Change in Serum Levels of IRT From Baseline Through | |
| | | Week 24 | |
| | 9.5.2.8 | Change in Microbiology Culture From Baseline at Week 24 | |
| | 9.5.2.9 | Absolute Change From Baseline in ppFEV1 at Week 24 | |
| | 9.5.2.10 | Absolute Change in Sweat Chloride From Week 24 at Week 26 | |
| | 9.5.2.11 | | |
| | 9.5.2.12 | $oldsymbol{\omega}$ | |
| | 9.5.2.13 | $oldsymbol{arepsilon}$ | |
| | | ves Listings | |
| 10 | | of Interim and IDMC Analyses | |
| | | Analysis | |
| | | Analysis | |
| 12 | | endices | |
| | | Schedule of Assessments | |
| | 1 1 | Analysis Visit Window Mapping Rules for Safety and Pharmacodynamic | |
| | | ements | |
| | 1 1 | Imputation Rules for Missing Prior/Concomitant Medication Dates | |
| | 1 1 | Imputation Rules for Missing AE dates | |
| | | Criteria for Potentially Clinically Significant Events | |
| | | Details of Statistical Methodology | 37 |
| | | Blood Pressure Normal Levels for Boys and Girls by Age and Height | 20 |
| | | ile | |
| | 1 1 | Important Protocol Deviation Programming Rules (Based on the Clinical | |
| | Databas | se) | 39 |



#### 4 INTRODUCTION

This statistical analysis plan (SAP) is for the final analysis of study VX15-809-115 Part B only and is based on the

- approved clinical study protocol, dated 13 April 2017, Version 3.0,
- approved eCRF, dated 16 December 2016, Version 4.0.

Study VX15-809-115 is a phase 3, 2-part, open-label study to evaluate the safety and pharmacokinetics (PK) of lumacaftor/ivacaftor combination therapy in subjects aged 2 through 5 years with cystic fibrosis, homozygous for the *F508del-CFTR* mutation.

This SAP (Methods) documents the planned final safety and pharmacodynamics analysis and data presentation for Part B of VX15-809-115.

SAS® Version 9.3 Software (SAS Institute, Cary, North Carolina, USA) or higher will be used to generate all statistical outputs (tables, figures, listings and datasets).

The SAP will be finalized and approved before the database lock for the final analysis for Part B. Any changes made to the SAP Methods after the above end of Part B activity has occurred will be documented in the clinical study report.

The analysis addressing the PK objective of the study will be described in the Clinical Pharmacology Analysis Plan (CPAP), which will be developed separately by the Clinical Pharmacology department at Vertex Pharmaceuticals Incorporated (Vertex).

### 5 STUDY OBJECTIVES

# 5.1 Primary Objective

#### Part A

To evaluate the PK of lumacaftor (LUM) and ivacaftor (IVA) and their respective metabolites in subjects aged 2 through 5 years with cystic fibrosis (CF), homozygous for F508del

#### Part B

To evaluate the safety of LUM/IVA combination therapy in subjects aged 2 through 5 years with CF, homozygous for *F508del* 

# 5.2 Secondary Objectives

#### Part A

To evaluate the safety of LUM/IVA combination therapy in subjects aged 2 through 5 years with CF, homozygous for *F508del* 

#### Part B

- To evaluate the pharmacodynamics (PD) of LUM/IVA combination therapy in subjects aged 2 through 5 years with CF, homozygous for *F508del*
- To evaluate the off-drug PD response after the Washout Period
- To evaluate the PK of LUM and IVA and their respective metabolites in subjects aged 2 through 5 years with CF, homozygous for *F508del*

# 5.3 Other Objectives

Not Applicable

#### 6 STUDY ENDPOINTS

# 6.1 Primary Endpoint

### Part A

PK parameters of LUM and IVA

#### Part B

Safety and tolerability assessments based on adverse events (AEs), clinical laboratory values (serum chemistry, hematology, coagulation studies, and urinalysis), standard 12-lead electrocardiograms (ECGs), vital signs, pulse oximetry, ophthalmological examinations, and spirometry

# 6.2 Secondary Endpoints

### Part A

- PK parameters of the metabolites of LUM and IVA
- Safety and tolerability assessments based on AEs, clinical laboratory values (serum chemistry, hematology, coagulation studies, and urinalysis), standard 12-lead ECGs, vital signs, pulse oximetry, and spirometry

#### Part B

- Absolute change from baseline in sweat chloride at Week 24
- Absolute change from baseline in body mass index (BMI) and BMI-for-age z-score at Week 24
- Absolute change from baseline in weight and weight-for-age z-score at Week 24
- Absolute change from baseline in stature and stature-for-age z-score at Week 24
- Time-to-first pulmonary exacerbation through Week 24
- Number of pulmonary exacerbations through Week 24
- Number of CF-related hospitalizations through Week 24

- Absolute change in fecal elastase-1 (FE-1) levels from baseline at Week 24
- Absolute change in serum levels of immunoreactive trypsinogen (IRT) from baseline through Week 24
- Change in microbiology cultures from baseline at Week 24
- Absolute change from baseline in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) at Week 24
- Absolute change in sweat chloride from Week 24 at Week 26
- Acceptability/palatability of LUM/IVA granules at Day 1
- Absolute change from baseline in lung clearance index (LCI)<sub>2.5</sub> at Week 24
- Absolute change from baseline in LCI<sub>5.0</sub> at Week 24
- PK parameters of LUM, IVA, and their respective metabolites

### 7 STUDY DESIGN

# 7.1 Overall Design

This is a Phase 3, 2-part, open-label, multicenter study evaluating the PK, safety, tolerability, and PD of multiple doses of LUM/IVA in subjects 2 through 5 years of age (inclusive) with CF, homozygous for *F508del*. Part A is designed to evaluate the PK of LUM and IVA and their respective metabolites and the safety of LUM/IVA combination therapy. Part B is designed to evaluate the safety and PD of LUM/IVA combination therapy and also to evaluate the PK of LUM and IVA and their respective metabolites.

Subjects who participate in Part A may participate in Part B, if they meet the eligibility criteria.

#### Part A

Approximately 12 subjects are planned for enrollment. Assuming a 10% dropout rate, approximately 10 subjects should complete Part A. Approximately half of the subjects should complete the study in each of the following weight groups: <14 kg and ≥14 kg at screening.

Part A includes the following:

- Screening Period (Day -28 through Day -1)
- Treatment Period (Day 1 through Day  $15 \pm 2$  days)
- Safety Follow-up Visit ( $10 \pm 3$  days after the last dose of LUM/IVA)

Figure 7-1 depicts the schematic for the Part A study design.

A review of safety, tolerability, and available PK data will be completed by an internal Vertex team after Part A to determine the dose(s) to be evaluated in Part B. Additional subjects or treatment cohorts may be enrolled, if data from the initial, planned, 12 subjects are inadequate to make a determination of the dose(s) to be evaluated in Part B.

Figure 7-1 Schematic of Study Design for Part A



IVA: ivacaftor; LUM: lumacaftor; q12h: every 12 hours

Notes: Approximately half of the subjects should complete the study in each of the following weight groups: <14 kg and ≥14 kg at screening. No dose adjustments will be made across the duration of study treatment. On Day 15, only the morning dose of LUM/IVA will be administered.

#### Part B

Approximately 56 subjects are planned for enrollment. Assuming a 10% dropout rate, approximately 50 subjects should complete Part B; at least 10 subjects must be <3 years of age at screening. Subjects should be ≥3 years of age at screening for enrollment in the optional LCI Substudy at a subset of sites. Additional subjects may be enrolled at the sponsor's discretion to achieve up to 30 subjects in the LCI Substudy.

Part B includes the following:

- Screening Period (Day -28 through Day -1)
- Treatment Period (Day 1 through Week  $24 \pm 5$  days)
- Washout Period (Week 24 to Week 26 ± 4 days)
- Safety Follow up Visit (Week 26 [2 weeks ± 4 days after the last study dose of LUM/IVA])

Figure 7-2 depicts the schematic for the Part B study design.

Subjects who have completed the required visits in Part B may be eligible to enroll in the Treatment Cohort or Observational Cohort of an Extension Study to evaluate long-term treatment with LUM/IVA; enrollment will be based on the eligibility criteria. The Treatment Cohort will enroll subjects who completed LUM/IVA treatment and the Safety Follow up Visit in Part B. The Observational Cohort will enroll subjects who received at least 4 weeks of LUM/IVA treatment in Part B and completed visits up to the Safety Follow up Visit, if applicable, in Part B, but do not meet eligibility criteria for enrollment into the Treatment Cohort. The Safety Follow up Visit, if applicable, is the last visit for Part B, and should also be the Day 1 Visit in the Extension Study.

In the later sections, all discussions and analyses plans will be limited to Part B only.

Figure 7-2 Schematic of Study Design for Part B



ETT: Early Termination of Treatment; IVA: ivacaftor; LCI: lung clearance index; LUM: lumacaftor; q12h: every 12 hours Notes: Approximately 56 subjects are planned for enrollment. Assuming a 10% dropout rate, approximately 50 subjects should complete Part B; at least 10 subjects must be <3 years of age. Subjects should be ≥3 years of age for enrollment in the optional LCI Substudy at a subset of sites. Additional subjects may be enrolled at the sponsor's discretion to achieve up to 30 subjects in the LCI Substudy.

- The doses listed above are the planned doses for Part B. Depending on the results from Part A, a single dose from Part A may be selected for all subjects in Part B or a previously unspecified dose or doses may be selected for Part B. No dose adjustments across the duration of treatment will be made. The last dose of LUM/IVA in Part B will be the evening dose before the Week 24 Visit.
- Subjects who prematurely discontinue LUM/IVA treatment will be asked to complete the ETT Visit, to remain on study, and to complete the study assessments from the time of LUM/IVA discontinuation through the Week 24 Visit and the Safety Follow-up Visit, if applicable. The Safety Follow-up Visit is not required for subjects who permanently discontinue LUM/IVA treatment before or at the Week 16 Visit if they return for the Week 24 Visit or for subjects who continue onto commercially-available LUM/IVA by prescription of a physician within 2 weeks (± 4 days) of completing LUM/IVA treatment at Week 24 or at the ETT Visit.
- Subjects who have completed the required visits in Part B may be eligible to enroll in the Treatment Cohort or Observational Cohort of an Extension Study to evaluate long-term treatment with LUM/IVA; enrollment will be based on the eligibility criteria.

#### Sample Size and Power

No formal sample size calculations have been performed. The number of subjects in Part B is deemed adequate to meet the primary safety objective. Given approximately 56 subjects are planned for enrollment and assuming a 10% dropout rate, approximately 50 subjects will complete Part B. Table 7-1 displays estimates of the probability for observing AEs in at least 1 subject for the given incidence ( $\theta$ ) and sample size. With a total sample size of 50 subjects (completers), there is a 92.3% chance of observing AEs in at least 1 subject if the true incidence is 5%, and a 99.5% chance of observing AEs in at least 1 subject if the true incidence is 10%. The probabilities are the binomial probabilities calculated using S-PLUS  $^{\otimes}$ .

Table 7-1 Probability of Observing Adverse Events in At Least 1 Subject if the Adverse Event Incidence (θ) is 5% and 10%

| Sample Size | $\theta = 5\%$ | $\theta = 10\%$ |
|-----------------|----------------|-----------------|
| 50 <sup>a</sup> | 92.3% | 99.5% |

<sup>50</sup> reflects the sample size of the completers.

Additional subjects may be enrolled at the sponsor's discretion to achieve up to 30 subjects in the LCI Substudy. This sample size is consistent with prior exploratory studies conducting LCI assessments.

### 7.2 Randomization

This is an open-label study with weight-based treatment group assignment. Randomization is not applicable.

# 7.3 Blinding and Unblinding

This is an open-label study. However for Part B, subjects and their legally appointed and authorized representative (e.g., parent or legal guardian) should not be informed of their study-related spirometry (subjects  $\geq 3$  years of age at screening), sweat chloride, and LCI results (subjects  $\geq 3$  years of age at screening who consent/assent to the optional LCI Substudy) during the study, regardless if the subject permanently discontinues treatment.

### 8 ANALYSIS SETS

# 8.1 All Subjects Set

All Subjects Set is defined as all subjects who have signed informed consent (and assent, if applicable) and enrolled, or dosed in Part B. This analysis set will be used for all individual subject data listings, unless specified otherwise.

# 8.2 Safety Set

Safety Set will include all subjects who received at least 1 dose of study drug in Part B. The Safety Set will be used for all safety analyses, with subjects analyzed according to the treatment they received, unless specified otherwise. In addition, the summary by the dosing groups (LUM 100 mg/IVA 125 mg q12h and LUM 150 mg/IVA 188 mg q12h) at enrollment determined by weight at the Screening Visit will be provided as supplementary information.

# 8.3 Full Analysis Set

Full Analysis Set (FAS) will include all enrolled subjects in Part B who are exposed to any amount of study drug in Part B. PD analyses (except LCI) will be based on the FAS.

# 8.4 LCI Substudy Set

LCI Substudy Set will include all subjects who have signed informed consent (and assent, if applicable) to the optional LCI Substudy in Part B and enrolled and dosed in Part B. LCI related analysis will be based on the LCI Substudy Set.
#### 9 STATISTICAL ANALYSIS

#### 9.1 General Considerations

The Part B Schedule of Assessments is provided in Appendix A. The precision standards for reporting safety variables are provided in an internal Biometrics document that specifies the programming rules including the precision for derived variables.

All individual subject data based on All Subjects Set will be presented in data listings.

Continuous variables will be summarized using the following descriptive summary statistics: number of subjects (n), mean, standard deviation (SD), standard error (SE), median, minimum (min), and maximum (max).

Categorical variables will be summarized using counts and percentages.

**Baseline value**, unless specified otherwise, will be defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of Part B study drug.

For ECGs, the Part B baseline value will be defined as the average of the pretreatment measurements on Day 1.

For LCI-related parameters, the values at each visit will be calculated from the technically acceptable washout replicates. The Part B baseline of LCI will be the most recent non-missing value calculated from the technically acceptable replicates before the initial administration of study drug.

For sweat chloride, the values at each visit will be based on the averaged measurements from left and right arms. The Part B baseline will be defined as the average of the values at screening of Part B and the pretreatment measurement on Day 1 of Part B. If only 1 pre-first dose measurement of sweat chloride is available, that measurement will be considered the Part B baseline.

**Change (absolute change) from baseline** will be calculated as postbaseline value - Part B baseline value.

**Relative change from baseline**: will be calculated and presented in percentage as  $100 \times (postbaseline \ value - \ Part \ B \ baseline \ value)/$  Part B baseline value.

**Treatment-emergent Period for Part B** will include the time period starting from the first dose date of the Part B study drug through 14 days after last dose of Part B study drug. The Treatment-Emergent period of Part B will be used for safety analyses unless specified otherwise.

**Unscheduled visits:** Unscheduled visit measurements will be included in analysis as follows:

- In scheduled visit windows per specified visit windowing rules
- In the derivation of baseline measurements/last on-treatment visit
- In the derivation of maximum/minimum values and maximum/minimum changes from baseline values
- In individual subject data listings as appropriate

**Visit windowing rules:** Appendix B defines the visit window mapping rules to derive the analysis visits for Part B.

Repeated observations within the same visits window:

- For all PD parameters, if there are multiple measurements within a visit window, the record at the scheduled visit will be used. If there are no measurements at the scheduled visit, then 1) the record closest to the target day will be used; or 2) if there are multiple records with the same distance to the target day, the latest record will be used.
- For all safety parameters, if there are multiple measurements within a visit window, then 1) the record closest to the target day will be used; or 2) if there are multiple records with the same distance to the target day, the latest record will be used.

BMI, weight, and stature will follow visit window rules for PD parameters when being considered as PD endpoints; they will follow visit window rules for safety parameters when being considered as safety endpoints. Their corresponding z-scores will be assigned analysis visit same as BMI, weight, and stature, respectively. Spirometry will follow the PD parameter window rule.

**Incomplete/missing data** will not be imputed, unless specified otherwise.

**Outliers:** No formal statistical analyses will be performed to detect or remedy the presence of statistical outliers, unless specified otherwise.

**Multiplicity:** No multiplicity adjustment will be performed and there is no hypothesis testing.

Unless otherwise specified, the analysis will be performed using descriptive summary statistics overall and by dosing groups (LUM 100 mg/IVA 125 mg q12h and LUM 150 mg/IVA 188 mg q12h). No statistical hypothesis testing will be performed.

#### 9.2 Background Characteristics

#### 9.2.1 Subject Disposition

The number of subjects in the following categories will be summarized overall and by dosing group:

- All Subjects Set
- Dosed (Safety Set)
- Enrolled and dosed (FAS)

The numbers and percentages (based on the Safety Set) of subjects in the following disposition categories will be summarized overall and by dosing group:

- Completed Part B study drug treatment
- Prematurely discontinued the Part B treatment
  - Reasons for discontinuations
  - Last completed scheduled on-treatment visit

- Completed Part B of study
- Prematurely discontinued the Part B of study and the reasons for discontinuations
- Rollover to extension study
  - Yes (Observational Cohort versus Treatment Cohort)
  - o No

The above disposition summary will also be provided based on the LCI Substudy Set.

A listing will be provided for subjects who discontinued Part B treatment or who discontinued Part B of study with reasons for discontinuation.

#### 9.2.2 Demographics and Baseline Characteristics

Demographics, medical history and baseline characteristics of Part B will be summarized overall and by dosing group based on the Safety Set.

Demographic data will include the following:

- Age at Part B baseline
- Age Group (< 3 and  $\ge 3$  years)
- Sex (female and male)
- Ethnicity (Hispanic or Latino, not Hispanic or Latino, and not collected per local regulations)
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Not Collected per Local Regulations and Other)

Baseline characteristics will include the following:

- Weight (kg)
- Weight Group ( $<14 \text{ kg and } \ge 14 \text{ kg}$ )
- Stature (cm)
- BMI (kg/m2)
- Weight-for-age z-score
- Stature-for-age z-score
- BMI-for-age z-score
- Sweat Chloride
- Spirometry (Subjects ≥3 years age at screening): FEV<sub>1</sub> (L), Percent Predicted FEV<sub>1</sub> (percentage points), FVC (L), Percent Predicted FVC(percentage points), FEF<sub>25-75%</sub> (L/s), Percent Predicted FEF<sub>25-75%</sub> (percentage points), FEV<sub>1</sub>/FVC, Percent Predicted FEV<sub>1</sub>/FVC (percentage points)

Similar tables for demographics and baseline characteristics will be provided based on the LCI Substudy Set. For that table, LCI<sub>2.5</sub> and LCI<sub>5.0</sub> summaries will also be summarized.

Medical history will be summarized by MedDRA system organ class (SOC) and preferred term (PT).

#### 9.2.3 Prior and Concomitant Medications

Medications used in this study will be coded by using the World Health Organization Drug Dictionary Enhanced (WHODDE) and categorized as the following:

- **Prior medication:** any medication that started before initial dosing of study drug in Part B, regardless of when it ended.
- Concomitant medication: medication continued or newly received at or after initial dosing of study drug in Part B to 14 days after the last dose of study drug in Part B.
- **Post-treatment medication:** medication continued or newly received after 14 days after the last dose of study drug in Part B.

A given medication can be classified as a prior medication, a concomitant medication, or a post-treatment medication; both prior and concomitant; both concomitant and post-treatment; or prior, concomitant, and post-treatment.

If a medication has a missing or partially missing start/end date or time and it cannot be determined whether it was taken before initial dosing, concomitantly, or after 14 days after the last dose of study drug, it will be considered as prior, concomitant, and post-treatment.

Prior medications and concomitant medications will be summarized descriptively by 1) preferred names; 2) anatomic class (ATC) level 1, ATC level 2, and preferred names based on the Safety Set.

Summaries of medications will be based on the Safety Set.

Details for imputing missing or partial start and/or stop dates of medication are described in Appendix C.

#### 9.2.4 Study Drug Exposure

Duration of Part B study drug exposure is defined as follows: Part B last dose date – Part B first dose date + 1 day, regardless of any interruptions in dosing. If the last dose date of Part B study drug is missing, the subject's last date in Part B will be used for analysis purposes.

Study drug exposure will be summarized descriptively (n, mean, SD, SE, median, min, and max in days) overall and by dosing group based on Safety Set.

Additionally, the cumulative duration of Part B treatment exposure, defined as the sum of the subject's duration of treatment exposure and expressed in subject-years, will be provided.

Duration of exposure will also be summarized as a categorical variable (>0 to  $\leq$ 2 weeks, >2 to  $\leq$ 4 weeks, >4 to  $\leq$ 8 weeks, >8 to  $\leq$ 16 weeks, >16 to  $\leq$ 24 weeks, and >24 weeks).

Exposure summaries will be based on the Safety Set.

#### 9.2.5 Study Drug Compliance

Part B study drug compliance will be assessed by calculating as follows:

 $100 \times (1 - [total number of days of Part B study drug interruption] / [duration of Part B study drug exposure + total number of days Part B study drug interrupted after last dose, if any]).$ 

The total number of days of study drug interruption is defined as the sum of (number of days of each study drug interruption), where number of days of each study drug interruption is defined as the interruption end date - the corresponding interruption start date + 1.

In calculating the total number of days of Part B study drug being interrupted, only the interruptions with duration of  $\geq 3$  days will be considered. An interruption with duration of  $\leq 3$  days will not be considered in the calculation.

Percent of stick packs taken will be calculated as follows:

 $100 \times (\text{total number of stick packs administered}) / (2 \times [\text{duration of study drug exposure in days} + \text{total number of days study drug interrupted after last dose, if any}]).$ 

Subjects who have a calculated percent of stick packs taken >100% will be considered as having taken 100% of stick packs.

Treatment compliance percentages and percent of stick packs taken will be summarized descriptively as quantitative variables (n, mean, SD, SE, median, minimum, and maximum) overall and by dosing group based on Safety Set. The number and percentage of subjects whose compliance is <80% or  $\ge80\%$  and the number and percentage of subjects whose percent of stick packs taken is <80% or  $\ge80\%$  will be summarized.

#### 9.2.6 Important Protocol Deviations

An important protocol deviation and violation (IPD) is a protocol deviation that has the potential to affect the interpretation of study results. IPD will be identified from the clinical database and/or site deviation log.

The rules for identifying important protocol deviations based on the clinical database are defined in Appendix H.

All IPDs will be presented in an individual subject data listing only.

#### 9.3 Efficacy Analysis

Not Applicable

#### 9.4 Safety Analysis

The overall safety profile of Part B study drug will be assessed in terms of the following safety and tolerability endpoints:

- Treatment-emergent adverse events (TEAEs)
- Clinical laboratory values (serum chemistry, hematology, coagulation studies, and urinalysis)
- ECGs (standard 12-lead)

- Vital signs
- Pulse oximetry
- Ophthalmological examinations
- Spirometry (Subjects ≥3 years age at screening)

Safety analyses will be performed overall and by dosing group. Safety analyses will be conducted for the Safety Set. Safety data will be presented in the individual subject data listings based on the All Subjects Set. Only descriptive summary statistics of safety data will be provided (i.e., no statistical hypothesis testing will be performed).

#### 9.4.1 Adverse Events

AEs will be classified as pretreatment AEs, TEAEs, or post-treatment AEs.

- **Pretreatment AE**: any AE that started before initial dosing of study drug in Part B.
- **TEAE**: any AE that increased in severity or that was newly developed during the Treatment Period which is defined as being the period from initial dosing of study drug in Part B to 14 days after the last dose of study drug in Part B.
- **Post-treatment AE**: any AE that increased in severity or that developed after 14 days after the last dose of study drug in Part B.

For AEs with missing or partial start dates, if there is no clear evidence that the AEs started before or after Part B study treatment, then the AEs will be classified as TEAEs for Part B.

Details for imputing missing or partial start dates of adverse events are described in Appendix D.

TEAE summaries will be presented using number and percentages of subjects.

An overview of TEAE profile will be provided, including total number of TEAEs, with number and percentage of subjects for the following categories: (1) All TEAEs, (2) Grades 3/4 TEAEs, (3) TEAEs by relationship to study drug, (4) TEAEs by maximum severity, (5) TEAEs leading to treatment interruption, (6) TEAEs leading to treatment discontinuation, (7) Serious TEAEs, (8) Serious TEAEs related to study drug, and (9) TEAEs leading to death.

AE summary tables will be presented for TEAEs only and will include the following:

- All TEAEs
- Grades 3/4 TEAEs
- TEAEs by relationship to study drug
- TEAEs by maximum severity
- TEAEs leading to treatment interruption
- TEAEs leading to treatment discontinuation
- Serious TEAEs

- Serious TEAEs related to study drug
- TEAEs leading to death
- Frequently reported TEAEs (≥5% at the preferred term level)

Summaries will be presented by MedDRA system organ class (SOC) and preferred term (PT) using frequency counts and percentages. When summarizing the number and percentage of subjects with an event, subjects with multiple occurrences of the same AE or a continuing AE will be counted once, only the maximum severity level will be presented in the severity summaries, and the worst/highest relationship level in the relationship summaries.

Separate tables will be provided summarizing the number of subjects, the number of events and the number of related events for the following by SOC and PT as per EudraCT requirement:

- Treatment-emergent Serious AEs
- Treatment-emergent Non-Serious AEs

#### Analysis of AEs of special interest (AESI) categories:

The following AESIs are defined:

1. Elevated Transaminases

The AESI of elevated transaminases is defined by the AEs whose PTs fall into any of the following:

- Alanine aminotransferase abnormal
- Alanine aminotransferase increased
- Aspartate aminotransferase abnormal
- Aspartate aminotransferase increased
- Transaminases abnormal
- Transaminases increased
- Liver function test abnormal
- Liver function test increased
- Hypertransaminasaemia
- Hepatic enzyme increased
- Hepatic enzyme abnormal
- 2. Respiratory Symptom AESI

The respiratory symptoms AESI is defined by the AEs whose PTs fall into any of the following:

Chest Discomfort

- Dyspnoea
- Respiration abnormal
- 3. Respiratory Event AESI (including respiratory symptoms or reactive airways)

The respiratory AESI of respiratory symptoms or reactive airways is defined by the AEs whose PTs fall into any of the following:

- Asthma
- Bronchial hyperreactivity
- Bronchospasm
- Chest Discomfort
- Dyspnoea
- Respiration abnormal
- Wheezing

Treatment-emergent AESIs will also be summarized

- 1. Showing number and percentage of subjects by PT;
- 2. Showing number and percentage of subjects by maximum severity;
- 3. Summary of duration of events (days) with descriptive statistics;
- 4. Summary of time-to-onset of the first event in days (relative to first dose date).
- 5. Showing number and percentage of subjects with TEAE leading to treatment discontinuation; with TEAE leading to treatment interruption; with serious TEAEs; with related serious TEAEs; and with TEAE leading to death.

In addition, listings that contain individual subject data for all TEAEs leading to treatment interruption, TEAEs leading to treatment discontinuation, deaths, and serious AEs will be provided separately. All AEs, including pre- and post-treatment AEs, will be presented in individual subject data listings.

#### 9.4.2 Clinical Laboratory

For laboratory measurements, the raw values and change from Part B baseline values of the continuous hematology/coagulation and chemistry results will be summarized overall and by dosing group in SI units at each scheduled time point. For hematology and chemistry, the number and percentage of subjects with abnormal low (<lower limit of normal [LLN]) value and with abnormal high (>ULN) value at each scheduled time point will be summarized.

The number and percentage of subjects with at least 1 categorical change during the Part B Treatment-Emergent period will be summarized. The categorical criteria are provided in Appendix E.

For each of the LFTs, mean (±SD) will be plotted at each timepoint.

Results of urinalysis will be listed in individual subject data listings only.

In addition, a listing containing individual subject hematology, chemistry, and coagulation values outside the normal reference ranges will be provided. This listing will include data from both scheduled and unscheduled visits.

#### 9.4.3 Electrocardiogram

For ECG measurements, a summary of raw values and change from Part B baseline values will be provided overall and by dosing group at each scheduled time point for the following standard 12-lead ECG measurements: RR (ms), HR (bpm), PR (ms), QRS duration (ms), QT (ms), and QT corrected for HR intervals [Fridericia's correction QTcF (ms) =QT/RR<sup>1/3</sup>]. In addition, the mean value at each time point will be plotted for QTcF.

The number and percentage of subjects with at least 1 categorical change during the Part B Treatment-Emergent period will be summarized. The categorical criteria are provided in Appendix E.

The number and percentage of subjects with shift changes from baseline (normal/missing, not clinically significant, and potentially clinically significant according to overall ECG evaluation) to the worst ECG evaluation during the Treatment Period will be summarized.

#### 9.4.4 Vital Signs

For vital signs measurements, the raw values and change from Part B baseline values will be summarized overall and by dosing group at each scheduled time point: systolic and diastolic blood pressure (mm Hg), body temperature (°C), pulse rate (beats per minute), and respiratory rate (breaths per minute).

In addition, respiratiory rate at each predose and the corresponding postdose timepoints will be summarized (1 hour, 2 hours, 4 hours, worse value of 1, 2 or 4 hours), absolute change from predose to the corresponding postdose (1 hour, 2 hours, 4 hours, worse value of 1, 2 or 4 hours) will also be summarized.

The number and percentage of subjects with at least 1 categorical change during the Treatment period will be summarized. The categorical criteria are provided in Appendix E.

Potentially abnormal SBP and DBP by their percentiles adjusted for sex, age and stature will be provided, including

- Number and percentage of subjects with categories  $\geq$ 90%-<95%,  $\geq$ 95%-<99% + 5 mmHg and  $\geq$ 99% + 5 mmHg)
- Number and percentage of subjects with SBP and DBP percentiles ≥95% once and twice during the treatment-emergent period will be provided.
- Number and percentage of subjects with SBP and DBP percentiles ≥95% at each visit will also be provided.

The stature adjustment will be based on stature-for-age z-scores and their corresponding percentiles using the standard normal distribution (Appendix G). The stature percentiles will be further mapped per the following rules:

Table 9-1 Grouped Percentiles for stature-for-age Z-scores

| Calculated Percentiles (%) | Grouped Percentiles (%) | |
|----------------------------|-------------------------|---|
| 0 – <7.5 | 5 | _ |
| 7.5 – <17.5 | 10 | |
| 17.5 – <37.5 | 25 | |
| 37.5 – <62.5 | 50 | |
| 62.5 – <82.5 | 75 | |
| 82.5 – < 92.5 | 90 | |
| 92.5 – 100 | 95 | |

The sex and age-adjusted normal range for SBP and DBP for each grouped stature percentiles is based on the SBP/DBP table in the National Heart, Lung, and Blood Institute (NHLBI) website (http://www.nhlbi.nih.gov/health-pro/guidelines/current/hypertension-pediatric-jnc-4/blood-pressure-tables).

#### 9.4.5 Pulse Oximetry

For the pulse oximetry measurements, a summary of raw values and change from Part B baseline values will be provided at each scheduled time point for the percent of oxygen saturation by pulse oximetry.

In addition, oxygen saturation at each predose and the corresponding postdose timepoints will be summarized (1 hour, 2 hours, 4 hours, worse value of 1, 2 or 4 hours), absolute change from predose to the corresponding postdose (1 hour, 2 hours, 4 hours, worse value of 1, 2 or 4 hours) will also be summarized.

The number and percentage of subjects with shift changes from Part B baseline (normal/missing and low according to the reference range) to the lowest percent of oxygen saturation during the Treatment Period will be provided.

## 9.4.6 Ophthalmological Examinations

Ophthalmological examination findings will be presented as a data listing.

## 9.4.7 Spirometry

Spirometry data will be summarized descriptively at each visit.

The following parameters of forced expiratory volume in 1 second (FEV<sub>1</sub> (L)) and percent predicted FEV<sub>1</sub> (ppFEV<sub>1</sub>), forced vital capacity (FVC) (L) and percent predicted FVC (ppFVC), FEV<sub>1</sub>/FVC (ratio) and ppFEV<sub>1</sub>/FVC as well as forced expiratory flow (FEF<sub>25%-75%</sub>) (L/s) and percent predicted FEF (ppFEF<sub>25%-75%</sub>) will be summarized using descriptive statistics<sup>1</sup>. The percent predicted values ppFEV<sub>1</sub>, ppFVC, ppFEV<sub>1</sub>/FVC and ppFEF<sub>25%-75%</sub> will be calculated using the standards of Global Lungs Initiative (GLI) as described in

Appendix F. In addition, the mean value (95% CI) at each time point will be plotted for the absolute change from Part B baseline in ppFEV<sub>1</sub>.

In addition, ppFEV1 at each predose and the corresponding postdose timepoints will be summarized (2 hours, 4 hours, worse value of 2 or 4 hours), absolute change from predose to the corresponding postdose (2 hours, 4 hours, worse value of 2 or 4 hours) will also be summarized.

In addition, a listing containing individual subject data will be provided.

#### 9.4.8 Physical Examination

Physical examination findings will be presented as a data listing only.

#### 9.4.9 Other Safety Analysis

Not applicable.

#### 9.5 Pharmacodynamic Analysis

PD analyses (except LCI) will be based on the FAS. LCI related analysis will be based on the LCI Substudy Set.

#### 9.5.1 Analysis of Primary Endpoints

Not applicable.

#### 9.5.2 Analysis of Secondary Pharmacodynamic Endpoints

### 9.5.2.1 Absolute Change From Baseline in Sweat Chloride at Week 24

For each subject and at each time point, 2 sweat chloride measurements will be collected: 1 from the right arm and 1 from the left arm. Of the 2 measurements, only the sweat chloride value obtained from a sample volume  $\geq 15~\mu L$  will be included in any analysis (i.e., a sample volume of 15  $\mu L$  is required for testing and therefore any samples with volumes <15  $\mu L$  will not be included in the analysis). The sweat chloride results for the left and right arms will be averaged and used in the analysis if the sweat chloride values for the left and right arms are both  $\geq 15~\mu L$ ; if only 1 arm is  $\geq 15~\mu L$ , then only that value will be used. Any sweat chloride values outside of the reportable range (i.e. <10 mmol/L or >160 mmol/L) will not be included in the analysis. If a subject has replicated measurements at a postbaseline time point, then the median of the values will be used in data analyses.

Descriptive summary statistics (n, mean, SD, SE, median, minimum, and maximum), along with the 95% confidence interval and within-group *P* value based on Normal approximation, will be provided for absolute change from baseline in sweat chloride at Week 24.

In addition, descriptive summary statistics, along with 95% confidence interval and withingroup *P* values based on Normal approximation, will be provided for all other visits. Mean (95% CI) at each visit, overall and by dosing groups will be plotted.

# 9.5.2.2 Absolute Change From Baseline in BMI/BMI-for-Age Z-score at Week 24

BMI z-score will be calculated by using Centers for Disease Control and Prevention (CDC) growth charts. The BMI z-score will be calculated as follows:

$$z = \begin{cases} \left(\frac{X}{M}\right)^{L} - 1 \\ LS \end{cases}, \quad L \neq 0$$

$$\frac{\ln\left(\frac{X}{M}\right)}{S} \quad , \quad L = 0$$

Where *X* is the derived BMI value in kg/m<sup>2</sup> based on the raw weight and raw height and *L*, *M*, and *S* are selected from the CDC BMI-for-age chart by subject sex and age. The BMIAGE file contains these parameters by sex (1=male, 2=female) and age; it is available at: http://www.cdc.gov/growthcharts/percentile\_data\_files.htm. Additionally, SAS code for calculating percentiles and z-scores is available at: http://www.cdc.gov/growthcharts/computer\_programs.htm.

NOTE: The CDC BMI-for-age charts are designed for use in pediatric populations (2 to 20 years of age).

Descriptive summary statistics (n, mean, SD, SE, median, minimum, and maximum), along with the 95% confidence interval and within-group *P* value based on Normal approximation, will be provided for absolute change from baseline in BMI and BMI-for-age z-score at Week 24.

In addition, descriptive summary statistics, along with 95% confidence interval and withingroup P values based on Normal approximation, will be provided at all other visits. Mean (95% CI) at each visit, overall and by dosing groups will be plotted.

# 9.5.2.3 Absolute Change From Baseline in Weight/Weight-for-Age Z-Score at Week 24

The calculation of weight z-score is similar to that of BMI z-score (using the CDC growth charts and the derivation described above). Using the same equation above, X in the equation is the collected weight and L, M, and S parameters are selected from the CDC weight-for-age chart. The WTAGE file contains these parameters by sex and age; it is available at the website <a href="http://www.cdc.gov/growthcharts/percentile\_data\_files.htm">http://www.cdc.gov/growthcharts/percentile\_data\_files.htm</a>.

NOTE: The CDC growth charts are designed for use in pediatric populations (2 to 20 years of age).

Descriptive summary statistics (n, mean, SD, SE, median, minimum, and maximum), along with 95% confidence interval and within-group *P* values based on Normal approximation, will be provided for absolute change from baseline in weight and weight-for-age z-score at Week 24.

In addition, descriptive summary statistics, along with 95% confidence interval and withingroup *P* values based on Normal approximation, will be provided at all other visits. Mean (95% CI) at each visit, overall and by dosing groups will be plotted.

# 9.5.2.4 Absolute Change From Baseline in Stature/Stature-for-Age Z-score at Week 24

The calculation of stature z-score is similar to that of BMI z-score (using the CDC growth charts and the derivation described above). Using the same equation above, X in the equation is the collected stature and L, M, and S parameters are selected from the CDC stature -for-age chart. The STATAGE file contains these parameters by sex and age; it is available at the website <a href="http://www.cdc.gov/growthcharts/percentile">http://www.cdc.gov/growthcharts/percentile</a> data files.htm.

NOTE: The CDC growth charts are designed for use in pediatric populations (2 to 20 years of age).

Descriptive summary statistics (n, mean, SD, SE, median, minimum, and maximum), along with 95% confidence interval and within-group *P* values based on Normal approximation, will be provided for absolute change from baseline in stature and stature-for-age z-score at Week 24.

In addition, descriptive summary statistics, along with 95% confidence interval and withingroup *P* values based on Normal approximation, will be provided at all other visits. Mean (95% CI) at each visit, overall and by dosing groups will be plotted.

# 9.5.2.5 Analysis of Pulmonary Exacerbation-related Other Secondary Pharmacodynamic Variables

- Time-to-first pulmonary exacerbation through Week 24: Time-to-first pulmonary exacerbation will be analyzed using Kaplan-Meier method. Cumulative incidence of pulmonary exacerbation will be summarized and plotted. Subjects without an exacerbation by Week 24 Visit will be censored at Week 24 Visit or at the last visit before the Safety Follow-up Visit for subjects with missing Week 24 Visit.
- Number of pulmonary exacerbations through Week 24: The number of pulmonary exacerbations through Week 24 [inclusive] (including both on-treatment events and events after treatment discontinuation), normalized by the time spent in the study (Week 24 date first dose date +1), will be summarized. For subjects with missing Week 24 visit, the last visit before Safety Follow-up Visit will be used instead of the Week 24 date.
- Number of CF-related hospitalizations through Week 24: For the number of CF-related hospitalizations through Week 24 [inclusive], the analysis will be similar to the analysis of the number of pulmonary exacerbations through Week 24.

#### 9.5.2.6 Absolute Change in FE-1 Levels From Baseline at Week 24

Descriptive summary statistics (n, mean, SD, SE, median, minimum, and maximum), along with 95% confidence interval and within-group *P* values based on Normal approximation, will be provided for absolute change from baseline in FE-1 levels at Week 24.

In addition, descriptive summary statistics, along with 95% confidence interval based on Normal approximation, will be provided at all other visits.

In addition, a summary of FE-1 values ( $<15 \mu g/g$  and  $>=15 \mu g/g$ ) shift from baseline to Week 24 will be displayed. A spaghetti plot of the FE-1 values will also be plotted.

Number and percentage of subjects with pancreatic insufficiency, defined as having FE-1 level  $<200 \mu g/g$ , will be provided at Week 24 and at baseline. The within-group shift will be tested based on McNemar's test.

# 9.5.2.7 Absolute Change in Serum Levels of IRT From Baseline Through Week 24

For each subject, the serum levels of IRT through Week 24 for each subject will be derived as the simple arithmetic mean at each visit (Day 15, Weeks 4, 8, 16, and 24), regardless of on-treatment measurement or measurement after treatment discontinuation. As long as there is at least 1 measurement available for a specific visit, the average of the corresponding visit will be calculated based on all available measurements. If all measurements are missing, then the average through Week 24 will be missing and the subject will not be included in the summary for the average through Week 24. The absolute change in serum levels of IRT from baseline through Week 24 will be derived similarly as the simple arithmetic mean of the absolute change in serum levels of IRT from baseline at each visit.

Summary statistics, along with 95% confidence interval and within-group P values based on Normal approximation, for absolute change from baseline in serum levels of IRT through Week 24 will be provided.

In additional, summary statistics, along with 95% confidence interval and within-group *P* values based on Normal approximation, will be provided at each visit.

In addition, a summary of IRT values (<14 ng/mL and >=14 ng/mL) shift from baseline to Week 24 will be displayed. A spaghetti plot of the IRT values will also be plotted.

## 9.5.2.8 Change in Microbiology Culture From Baseline at Week 24

The presence of bacteria will be descriptively summarized by subject counts and percentages by visit and dosing group.

## 9.5.2.9 Absolute Change From Baseline in ppFEV1 at Week 24

Summary statistics, along with 95% confidence interval and within-group P values based on Normal approximation, for absolute change from baseline in ppFEV<sub>1</sub> will be provided at Week 24 [1].

In addition, summary statistics, along with 95% confidence interval and within-group *P* values based on Normal approximation, will be provided at all other visits. Mean (95% CI) at each visit, overall and by dosing groups will be plotted.

#### 9.5.2.10 Absolute Change in Sweat Chloride From Week 24 at Week 26

Summary statistics, along with 95% CI and within-group *P* values based on Normal approximation, for absolute change from Week 24 will be provided at Week 26.

#### 9.5.2.11 Acceptability/Palatability of LUM/IVA Granules at Day 1

Summary statistics will be provided for the acceptability/palatability data.

#### 9.5.2.12 Absolute Change From Baseline in LCI2.5 at Week 24

The LCI assessment at scheduled visits will be performed in multiple replicates. The LCI values at each visit included in the analysis will be the value calculated from the technically acceptable washout replicates.

When there is only one LCI value considered acceptable by the LCI central reader, the value will NOT be used. The assessment for that subject at the corresponding visit will not be included in the analysis; when there are at least 2 LCI values considered acceptable by the LCI central reader, the arithmetic mean of the values from the accepted trials will be calculated as the value at the corresponding visit.

Descriptive summary statistics (n, mean, SD, SE, median, minimum, and maximum), along with 95% confidence interval and within-group *P* values based on Normal approximation, will be provided for absolute change from baseline in LCI<sub>2.5</sub> at Week 24.

In addition, descriptive summary statistics, along with 95% confidence interval and withingroup *P* values based on Normal approximation, will be provided at all other visits. Mean (95% CI) at each visit, overall and by dosing groups will be plotted.

#### 9.5.2.13 Absolute Change From Baseline in LCI5.0 at Week 24

Analysis of absolute change in LCI<sub>5.0</sub> from baseline at Week 24 will be similar to the analysis of absolute change in LCI<sub>2.5</sub> from baseline at Week 24.

#### 9.6 Narratives Listings

Narratives listings will be provided for subjects with any of the following events that occurred by the study cutoff date:

- Death
- Serious AEs
- TEAEs leading to treatment discontinuation
- LFT elevations meeting at least 1 of the following criteria:
  - o ALT or AST > 5xULN, or
  - o ALT>3xULN and total bilirubin>2xULN, or
  - AST>3xULN and total bilirubin>2xULN

during the treatment-emergent period

#### 10 SUMMARY OF INTERIM AND IDMC ANALYSES

#### 10.1 Interim Analysis

Details of the Interim Analysis (IA) analysis will be provided in the IA/DMC Analysis Plan.

#### 10.2 IDMC Analysis

Details of the IDMC (Section 8.2 of the protocol) analysis will be provided in the IA/DMC Analysis Plan.

#### 11 REFERENCES

<sup>1</sup>Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall G, Culver BH, et al. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012;40(6):1324-43.

#### 12 LIST OF APPENDICES

**Appendix A: Schedule of Assessments** 

Table 12-1 Study VX15-809-115: Part B Screening

| Assessment | Screening Visit Day -28 through Day -1 |
|---|---|
| Informed consent/assent | X |
| Demographics | X |
| Medical and ophthalmological history | X |
| Stature, weight, and vital signs <sup>a,b</sup> | X |
| Pulse oximetry <sup>b</sup> | X |
| Ophthalmologic examination <sup>c</sup> | X |
| Full physical examination | X |
| Standard 12-lead ECG <sup>d</sup> | X |
| CFTR genotype <sup>e</sup> | X |
| Serum chemistry <sup>f</sup> | X |
| Hematology <sup>f</sup> | X |
| Coagulation studies <sup>f</sup> | X |
| Urinalysis <sup>f</sup> | X |
| Sweat chloride <sup>g</sup> | X |
| LCI (optional) <sup>h</sup> | X |
| Spirometry <sup>i</sup> | X |
| Medications review <sup>j</sup> | Continuous from signing of ICF through Safety Follow-up Visit (if required) |
| Adverse events | Continuous from signing of ICF through Safety Follow-up Visit (if required) |

BMI: body mass index; CFTR: cystic fibrosis transmembrane conductance regulator gene; ECG: electrocardiogram; ICF: informed consent form; LCI: lung clearance index

If children can stand unassisted and follow directions, stature should be measured as height; otherwise, stature will be measured as length. Stature and weight must be measured with shoes off and while wearing light clothing. BMI will be derived from this assessment. Refer to Section 11.4.3 of the protocol for details.

The subject should rest for at least 5 minutes before having vital signs and pulse oximetry measured. Refer to Section 11.6.4 of the protocol for details.

An ophthalmologic examination will be conducted by a licensed ophthalmologist. The examination does not need to be repeated if there is documentation of an examination meeting protocol criteria that was conducted within 3 months before the Screening Visit. Subjects with documentation of bilateral lens removal do not need the ophthalmologic examination. Refer to Section 11.6.6 of the protocol for details.

A standard 12-lead ECG will be performed. The subject will be instructed to rest in the supine position for at least 5 minutes, if possible, before having an ECG performed. The ECG will be performed before any other procedures that may affect heart rate, such as blood draws. Refer to Section 11.6.5 of the protocol for details.

All subjects will be tested to assess *CFTR* genotype, regardless of availability of a previous *CFTR* genotype laboratory report. Refer to Section 11.6.2 of the protocol for details. However, this assessment does not need to be repeated for confirmed subjects in Part A who may participate in Part B.

Refer to Section 11.6.2 of the protool for details.

If an eligible historical sweat chloride result is documented in the subject's medical record, that result alone (and not the Screening Visit result) may be used to determine eligibility. For subjects using an historical sweat chloride value documented in their medical record to determine eligibility, the sweat chloride test at the Screening Visit is still required. At screening, 2 samples may be collected, 1 sample from each arm (left and right).

h The LCI assessment (subjects ≥3 years of age at screening who consent/assent to the optional LCI Substudy) may be performed pre- or post-bronchodilator. The assessment will be performed in multiple replicates and before the spirometry assessment. Refer to Section 11.4.2 of the protocol for details.

<sup>&</sup>lt;sup>i</sup> Spirometry (subjects ≥3 years of age at screening only) may be performed pre- or post-bronchodilator. Refer to Section 11.6.7 of the protocol for details.

Refer to Section 9.4.2 of the protocol for details.

| + |
|-----------------|
| Visi |
| Follow-up |
| etv |
| Safet |
| SP |
| an |
| po |
| t Period |
| t P |
| reatmen |
| Ε |
| B |
| Part |
| 3 |
| = |
| 60 |
| 5-8 |
| dv VX15-809-115 |
| A |
| Stu |
| 2-2 |
| e 1 |
| abl |

| 00000 | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Treatment Period | Period | | | | | Safety |
| | | | | | | | | | | | Follow-up Visit |
| | | | | | | | | | | | (Week 26 |
| | | | | | | | | | | Early | [2 weeks |
| | | Day 3 | | | | | | | | Termination | ± 4 days |
| | Day 1 | (± 1 | Day 15 | Week 4 | Week 8 | Week 12 | Week 16 Week 20 | | Week 24 | Week 24 of Treatment | After Last |
| Event/Assessment <sup>a</sup> | 22 | day) | | | (± 5 days) | $(\pm 5 \text{ days}) \mid (\pm 5 \text{ days}) \mid (\pm 5 \text{ days}) \mid (\pm 5 \text{ days}) \mid (\pm 5 \text{ days}) \mid (\pm 5 \text{ days})$ | (± 5 days) | (± 5 days) | (± 5 days) | (ETT) Visit <sup>b</sup> | Dose]) <sup>c,d</sup> |
| Clinic visit | X | | X | X | X | | X | | X | X | X |
| Telephone contacte | | X | | | | X | | X | | | |
| Stature and weight <sup>f</sup> | X | | X | X | X | | X | | X | X | X |
| Vital signs <sup>g</sup> | $X_{ m p}$ | | X | X | X | | X | | X | X | X |
| Pulse oximetry <sup>g</sup> | X | | X | X | X | | X | | X | X | X |
| Ophthalmologic examination | | | | | | | | | $X^{i}$ | $X^{i}$ | X |

All assessments will be performed before LUM/IVA dosing unless noted otherwise (Section 11.1 of the protocol). When repeats of an assessment are required postdose at a given visit, the assessment will be collected only once if LUMIVA is not administered on the day of the visit (i.e., LUMIVA interruption or permanent LUMIVA

time of LUM/IVA treatment discontinuation through the Week 24 Visit and Safety Follow-up Visit, if applicable. The ETT Visit should be scheduled as soon as possible Subjects who prematurely discontinue LUM/TVA treatment will be asked to complete the ETT Visit, to remain on study, and to complete the study assessments from the become eligible to receive commercially-available LUM/IVA by prescription of a physician, and who choose to continue onto commercially-available LUM/IVA before after the subject decides to terminate LUM/IVA treatment. If the ETT Visit occurs 10 days or later following the last dose of LUM/IVA, then the ETT Visit will replace the Safety Follow-up Visit (i.e., the assessments performed will be those specified for the ETT Visit), and a Safety Follow-up Visit will not be required. Subjects who completion of Part B, must remain on study-supplied LUM/IVA through the ETT Visit, and may only initiate treatment with commercially-available LUM/IVA after completion of this visit.

The Safety Follow-up Visit is not required for subjects who permanently discontinue LUM/TVA treatment before or at the Week 16 Visit if they return for the Week 24 Visit. The Safety Follow-up Visit is not required for subjects who continue onto commercially-available LUMIVA by prescription of a physician within 2 weeks (± 4 days) of completing LUM/IVA treatment at Week 24 or at the ETT Visit.

The Safety Follow-up Visit, if applicable, is the last visit for Part B, and should also be the Day 1 Visit in the Extension Study (refer to Section 8.1.2 of the protocol and the Extension Study for details)

Telephone contacts will be made to assess the subject's status, any AEs, concomitant medications, treatments, and procedures.

If children can stand unassisted and follow directions, stature should be measured as height; otherwise, stature will be measured as length. Stature and weight must be measured with shoes off and while wearing light clothing. BMI will be derived from this assessment. Refer to Section 11.4.3 of the protocol for details.

The subject should rest for at least 5 minutes before having vital signs and pulse oximetry measured. Refer to Section 11.6.4 of the protocol for details.

An ophthalmologic examination will be conducted by a licensed ophthalmologist at the Week 24 Visit OR the Safety Follow-up Visit OR the ETT Visit, as applicable. Subjects with documentation of bilateral lens removal do not need the ophthalmologic examination. Refer to Section 11.6.6 of the protocol for details. Vital signs will be measured predose and at 1 hour (± 15 minutes), 2 hours (± 15 minutes), and 4 hours (± 15 minutes) postdose on Day 1.

Study VX15-809-115: Part B Treatment Period and Safety Follow-up Visit **Table 12-2** 

| | | | | | Treatment Period | Period | | | | | Safety |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day 3 | | | | | | | | Early<br>Termination | Follow-up Visit<br>(Week 26<br>[2 weeks<br>± 4 days |
| Event/Assessment <sup>a</sup> | Day 1 | (± 1<br>day) | Day 15<br>(± 3 days) | Week 4 (± 5 days) | Week 8<br>(± 5 days) | Week 12 (± 5 days) | Week 16<br>(± 5 days) | Week 20 (± 5 days) | Week 24 (± 5 days) | of Treatment<br>(ETT) Visit <sup>b</sup> | After Last<br>Dose]) <sup>c,d</sup> |
| Full physical examination | X | | | | | | | | X | X | X |
| Abbreviated physical examination | $X_k$ | | | | | | | | | | |
| Standard 12-lead ECG <sup>1</sup> | $X_{m}$ | | X | X | X | | X | | X | X | X |
| Serum chemistry <sup>n</sup> | X | | X | X | X | | X | | X | X | X |
| Hematology <sup>n</sup> | | | X | X | X | | X | | X | X | |
| Coagulation studies <sup>n</sup> | | | | | | | | | X | X | |
| Urinalysis <sup>n</sup> | X | | | | | | | | X | X | X |
| Qualitative microbiology cultures° | X | | | | | | | | X | | |
| PK sampling <sup>p</sup> | | | X | X | | | | | X | | |
| Immunoreactive trypsinogen | X | | X | X | X | | X | | X | X | X |
| Fecal elastase-1 <sup>q</sup> | X | | X | X | X | | X | | X | X | X |
| Sweat chloride <sup>r</sup> | X | | | X | | | | | X | X | X |

Symptom-directed physical examinations will occur at any time during the study if triggered by AEs or if deemed necessary by the investigator. Refer to Section 11.6.4 of the protocol for details.

An abbreviated physical examination will be performed 4 hours (# 30 minutes) postdose on Day 1. Refer to Section 11.6.4 of the protocol for details.

performed. The ECG will be performed before any other procedures that may affect heart rate, such as blood draws. Refer to Section 11.6.5 of the protocol for details. A standard 12-lead ECG will be performed. The subject will be instructed to rest in the supine position for at least 5 minutes, if possible, before having an ECG

Standard 12-lead ECGs will be performed predose and at 4 hours (± 15 minutes) postdose on Day 1. Predose ECGs on Day 1 will be performed in triplicate.

<sup>n</sup> Refer to Section 11.6.2 of the protocol for details.

Refer to Section 11.4.7 of the protocol for details.

At the Day 15 and Week 4 Visits, PK blood samples will be collected predose (within 60 minutes before dosing) and 2 to 6 hours after the morning dose. At the Week 24 Visit, PK blood samples will be collected at the same time as other blood collections. Refer to Section 11.3.1 of the protocol for details.

Samples will be collected at the study center during the study visit; however, samples may be collected by the subject's caregiver up to 24 hours before the study visit (Section 11.4.5 of the protocol). The sample may be collected pre- or postdose.

The sweat chloride test must be conducted predose relative to the morning dose of LUM/IVA during the Treatment Period (at approximately the same time as predose blood collections). At each time point, 2 samples will be collected, 1 sample from each arm (left and right). Refer to Section 11.4.1 of the protocol for details.

Vertex Pharmaceuticals Incorporated

Study VX15-809-115: Part B Treatment Period and Safety Follow-up Visit **Table 12-2** 

| | | | | | Treatment Period | Period | | | | | Safety |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | Follow-up Visit<br>(Week 26 |
| | | | | | | | | | | Early | [2 weeks |
| | | Day 3 | | | | | | | | Termination | ± 4 days |
| | Day 1 | (± 1 | Day 15 | Week 4 | Week 8 | Week 12 | Week 16 | Week 20 | Week 24 | of Treatment | After Last |
| Event/Assessment <sup>a</sup> | 122 | day) | (± 3 days) | (± 5 days) | (± 5 days) | (± 5 days) | (± 5 days) | (± 5 days) | (± 5 days) | (ETT) Visit <sup>b</sup> | Dose]) <sup>c,d</sup> |
| LCI (optional) <sup>\$</sup> | X | | | X | | | | | X | X | X |
| Spirometry <sup>t</sup> | $\mathbf{X}_{\mathbf{n}}$ | | X | X | X | | X | | X | X | X |
| Other events related to | X | | X | X | X | X | X | X | X | X | |
| outcome | | | | | | | | | | | |
| LUM/IVA dosing <sup>w</sup> | | | | | LUM/IVA q12h | q12h | | | | | |
| Observation 4 hours after the | X | | | | | | | | | | |
| first dose | | | | | | | | | | | |
| Acceptability/palatability | X | | | | | | | | | | |
| assessment | | | | | | | | | | | |
| Study drug count | | | X | X | X | | X | | X | X | |
| Medications, treatments, and procedures review <sup>y</sup> | | | | Continuor | ıs from signii | Continuous from signing of ICF through Safety Follow-up Visit (if required) | ough Safety I | ollow-up Vi | sit (if require | (pa | |
| Adverse events | | | | Continuor | 15 from signii | Continuous from signing of ICF through Safety Follow-up Visit (if required) | ough Safety I | ollow-up Vi | sit (if require | (pa | |
| AE: adverse event: BMI: body mass index: CF: cystic fibrosis: ECG: electrocardiogram: ETT: Early Termination of Treatment: ICF: informed consent form: IVA: ivacaftor: | nass inde | x: CF: cv | vstic fibrosis: | FCG: electro | cardiogram: | FTT: Early | Termination of | of Treatment | ICF: inform | ed consent form | . IVA: ivacaftor: |

LCI: lung clearance index; LUM: lumacaftor; PK: pharmacokinetic; q12h: every 12 hours

The LCI assessment (subjects  $\ge$  years of age at screening who consent/assent to the optional LCI Substudy) should be performed pre-bronchodilator and before

LUMIVA dosing (Section 11.4.2 of the protocol). The assessment will be performed in multiple replicates and before the spirometry assessment. Spirometry (subjects  $\ge$  3 years of age at screening only) should be performed pre-bronchodilator. Refer to Section 11.6.7 of the protocol for details.

Other events related to outcome include assessments relating to pulmonary exacerbations, administration of antibiotic therapy for sinopulmonary signs or symptoms, and Day 1 spirometry will be performed before LUM/IVA dosing and at 2 hours ( $\pm$  30 minutes) and 4 hours ( $\pm$  30 minutes) postdose.

<sup>(</sup>Section10.2 of the protocol). On days of scheduled visits, the morning dose of LUM/IVA will be administered at the site after predose assessments have been completed. At the Week 24 Visit, the morning dose of LUM/IVA will NOT be administered. The last dose of LUM/IVA in Part B will be the evening dose administered LUMIVA will be administered q12h (± 2 hours) within 30 minutes of consuming fat-containing food such as a standard CF high-fat, high-calorie meal or snack hospitalizations (Section 11.4.4 of the protocol).

Refer to Section 11.4.9 of the protocol for details. Refer to Section 9.4.2 of the protocol for details. the day before the Week 24 Visit.

# Appendix B: Analysis Visit Window Mapping Rules for Safety and Pharmacodynamic Measurements

Table 12-3 Visit Window Mapping Rules for Safety and Pharmacodynamic Measurements

| Assessments | Visit | Target Study Day | Visit Window (in study days) |
|---|---|---|---|
| Spirometry | Day 15 | 15 | (1, 22] |
| <ul> <li>Weight and stature</li> </ul> | Week 4 | 29 | [23, 43] |
| • Labs | Week 8 | 57 | [44, 85] |
| <ul> <li>Chemistry</li> </ul> | Week 16 | 113 | [86, 141] |
| <ul> <li>Hematology</li> </ul> | Week 24 | 169 | [142, 176] |
| <ul> <li>Vital signs</li> </ul> | | | |
| <ul> <li>Pulse oximetry</li> </ul> | | | |
| <ul> <li>Standard digital ECG</li> </ul> | | | |
| • Fecal elastase -1 | | | |
| • Immunoreactive trypsinogen | | | |
| • Labs | Week 24 | 169 | (1, 176] |
| <ul> <li>Coagulation</li> </ul> | | | - |
| • Ophthalmologic exam | | | |
| Sweat chloride | Week 4 | 29 | (1, 99] |
| • LCI | Week 24 | 169 | [100, 176] |

# Special handling for Spirometry (for the change from predose to postdose analysis only):

For the change from predose to postdose spirometry analysis only, no windowing rules are used.

- 1. Predose spirometry: analysis visit = nominal visit;
- 2. Postdose 2-hour/4-hour spirometry: analysis visit = nominal visit.

# **Special handling for VS/ECG (for the change from predose to postdose analysis only):** For the change from predose to postdose VS/ECG analysis only, no windowing rules are used.

- 1. Day 1 predose VS/ECG: analysis visit = nominal visit for Day 1, Predose.
- 2. Day 1 post-dose VS/ECG by hour: analysis visit = nominal visit.

#### **Special handling for Follow-up:**

Follow-up will use the nominal visit and will not follow the visit window rule.

#### **Appendix C: Imputation Rules for Missing Prior/Concomitant Medication Dates**

Imputation rules for missing or partial medication start/stop dates are defined below:

- 1. Missing or partial medication start date:
  - a. If only DAY is missing, use the first day of the month.
  - b. If DAY and Month are both missing, use the first day of the year.
  - c. If DAY, Month and Year are all missing, use a date before the first dose date.
- 2. Missing or partial medication stop date:
  - a. If only DAY is missing, use the last day of the month.
  - b. If DAY and Month are both missing, use the last day of the year.
  - c. If DAY, Month and year are all missing, assign 'continuing' status to stop date.

In summary, the prior, concomitant or post categorization of a medication is described below.

Table 12-4 Prior, Concomitant, and Post Categorization of a Medication

| Medication Start Date | Study Drug | Medication Stop Date ≥ First Dose Date and ≤ End Date of Treatment-emergent Period | > End Date of<br>Treatment-emergent<br>Period |
|---|---|---|---|
| | P | PC | PCA |
| < First dose date of study drug | F | PC | PCA |
| ≥ First dose date and | - | С | CA |
| ≤ End date of Treatment- | | | |
| emergent period | | | |
| > End date of Treatment- | - | - | A |
| emergent period | | | |

A: Post; C: Concomitant; P: Prior

#### **Appendix D: Imputation Rules for Missing AE dates**

Imputation rules for missing or partial AE start date are defined below:

#### If only Day of AE start date is missing:

If the AE start year and month are the same as that for the first dose date, then:

- If the full (or partial) AE end date is NOT before the first dose date or AE end date is missing, then impute the AE start day as the day of first dose date; otherwise, impute the AE start day as 1.
- Otherwise, impute the AE start day as 1.

Compare the imputed AE start date with Treatment-Emergent period to determine whether the AE is pretreatment AE, TEAE or post-treatment AE.

#### If Day and Month of AE start date are missing:

If AE start year = first dose year, then:

- If the full (or partial) AE end date is NOT before the first dose date or AE end date is missing, then impute the AE start Month and Day as the Month and Day of first dose date; otherwise, impute the AE start Month as January and the Day as 1.
- Otherwise, impute the AE start MONTH as January and the DAY as 1.

Compare the imputed AE start date with Treatment-Emergent period to determine whether the AE is pretreatment AE, TEAE or post-treatment AE.

#### If Year of AE start date is missing:

If the year of AE start is missing or AE start date is completely missing then query site with no imputation. Also compare the full (or partial) AE end date to the first dose date. If the AE end date is before the first dose date then the AE should be considered as a pretreatment AE. Otherwise, the AE will be considered as TEAE.

## **Appendix E: Criteria for Potentially Clinically Significant Events**

 Table 12-5
 Criteria for Potentially Clinically Significant Laboratory Tests

| Parameter | Categorical change | Comments |
|---|---|---|
| Clinical Chemistry | y | |
| ALT | ≤3xULN*(Not a categorical change) >3x - ≤ 5xULN >5x - ≤ 8xULN >3xULN >5xULN >8xULN | FDA DILI Guidance Jul 2009. |
| AST | ≤3xULN*( Not a categorical change) >3x - ≤ 5xULN >5x - ≤ 8xULN >3xULN >5xULN >8xULN | FDA DILI Guidance Jul 2009. |
| ALT or AST | ALT>3xULN or AST>3xULN | Vertex LFT working group 2014 |
| ALT or AST | ALT>5xULN or AST>5xULN | |
| ALT or AST | ALT>8xULN or AST>8xULN | |
| Alkaline<br>Phosphatase | >1.5xULN | FDA DILI Guidance Jul 2009. |
| Total Bilirubin | >1.5x - ≤2xULN<br>>2xULN | FDA DILI Guidance Jul 2009. |
| ALT and Total<br>Bilirubin | ALT>3xULN and TBILI>2xULN | FDA DILI Guidance Jul 2009. To be counted within a same treatment phase, whatever the interval between measurements. |
| AST and Total<br>Bilirubin | AST>3xULN and TBILI>2xULN | FDA DILI Guidance Jul 2009. To be counted within a same treatment phase, whatever the interval between measurements. |
| (ALT or AST) and<br>Total Bilirubin | (ALT>3xULN or AST>3xULN) and TBILI>2×ULN | Vertex LFT working group 2014 |
| СРК | $>3x - \le 10xULN$<br>>10xULN | FDA criteria Feb 2005.<br>Am J Cardiol April 2006. |
| Creatinine | ≥150 µmol/L (Adults)<br>≥30% change from baseline<br>≥100% change from baseline | Benichou C., 1994. |
| Blood Urea<br>Nitrogen | ≥17 mmol/L | |
| Chloride | <85 mmol/L<br>>115 mmol/L | |
| Sodium | $\leq$ 129 mmol/L $\geq$ 150 mmol/L | |

Table 12-5 Criteria for Potentially Clinically Significant Laboratory Tests

| Parameter | Categorical change | Comments |
|---|---|---|
| Potassium | <3 mmol/L<br>≥5.5 mmol/L | FDA Feb 2005. |
| Glucose | | |
| Hypoglycaemia | ≤3.9 mmol/L and <lln< td=""><td>ADA May 2005.</td></lln<> | ADA May 2005. |
| Hyperglycaemia | $\geq$ 11.1 mmol/L (unfasted); $\geq$ 7 mmol/L (fasted) | ADA Jan 2008. |
| Albumin | ≤25 g/L | |
| Hematology | | |
| WBC | <3.0 Giga/L (Non-Black); <2.0 Giga/L (Black)<br>≥16.0 Giga/L | Increase in WBC: not relevant. To be interpreted only if no differential count available. |
| Lymphocytes | >4.0 Giga/L | |
| Neutrophils | <1.5 Giga/L (Non-Black);<1.0 Giga/L (Black) | International Consensus meeting on drug-<br>induced blood cytopenias, 1991.<br>FDA criteria. |
| Monocytes | >0.7 Giga/L | |
| Basophils | >0.1 Giga/L | |
| Eosinophils | >0.5 Giga/L or >ULN (if ULN≥0.5 Giga/L) | Harrison- Principles of internal Medicine 17th Ed., 2008. |
| Hemoglobin | ≤115 g/L (Male); ≤95 g/L (Female)<br>≥185 g/L (Male); ≥165 g/L (Female) | Criteria based upon decrease from baseline are more relevant than based on absolute value. Other categories for decrease from |
| | Decrease from Baseline ≥20 g/L | baseline can be used ( $\geq$ 30 g/L, $\geq$ 40 g/L, $\geq$ 50 g/L). |
| Hematocrit | ≤0.37 v/v (Male) ; ≤0.32 v/v (Female)<br>≥0.55 v/v (Male) ; ≥0.5 v/v (Female) | |
| RBC | ≥6 Tera/L | |
| Platelets | <100 Giga/L<br>≥700 Giga/L | International Consensus meeting on drug-<br>induced blood cytopenias, 1991. |

Table 12-6 Criteria for Potentially Clinically Significant ECGs

| Parameter | Categorical change | Comments |
|-----------|---------------------------------------------|----------|
| HR | ≤50 bpm and decrease from baseline ≥20 bpm | |
| | ≥120 bpm and increase from baseline ≥20 bpm | 1 |
| | <40 bpm | |
| | <50 bpm | |
| | >90 bpm | |
| PR | ≥220 ms and increase from baseline ≥20 ms | |

Table 12-6 Criteria for Potentially Clinically Significant ECGs

| Parameter | Categorical change | Comments |
|---|---|---|
| QRS | ≥120 ms | |
| QTc<br>Borderline<br>Prolonged*<br>Additional | Absolute values (ms) Borderline: 431-450 ms (Male); 451-470 ms (Female) Prolonged: >450 ms (Male); >470 ms (Female) ≥500 ms | To be applied to any kind of QT correction formula. |
| | Increase from baseline Borderline: Increase from baseline 30-60 ms Prolonged: Increase from baseline >60 ms | |

Note: Based on CPMP 1997 guideline.

Table 12-7 Criteria for Potentially Clinically Significant Vital Signs

| Parameter | Categorical change | Comments |
|---|---|---|
| Pulse Rate | ≤50 bpm and decrease from baseline ≥20 bpm ≥120 bpm and increase from baseline≥20 bpm | To be applied for all positions (including missing) except STANDING. |
| Weight | ≥5% increase from baseline<br>≥5% decrease from baseline | FDA criteria Feb 2007. |

#### Appendix F: Details of Statistical Methodology

Percent predicted values will be calculated for parameters of FEV<sub>1</sub>, FVC, FEV1/FVC, and FEF<sub>25%-75%</sub> using the Quanjer GLI-2012 Regression Equations and Lookup Tables.

The regression equations and lookup tables required to implement the Quanjer GLI-2012 predicted values are available in:

Quanjer GLI-2012 Regression Equations and Lookup Tables. Philip H. Quanjer, Sanja Stanojevic, Tim J. Cole, Janet Stocks. Version 7 April 2013. Available at: http://www.erseducation.org/guidelines/global-lung-function-initiative/tools/quanjer-gli-2012-regression-equations-and-lookup-tables.aspx. Accessed 08 December 2015.

The instructions and tools on how to implement the Quanjer GLI-2012 equations are:

Implementing GLI-2012 regression equations. Philip H. Quanjer, Sanja Stanojevic, Tim J. Cole, Janet Stocks. Version 19 July 2015. Available at: http://www.erseducation.org/guidelines/global-lung-function-initiative/gli-2012-explained.aspx. Accessed 08 December 2015.

GLI-2012 - SAS Macro. Sanja Stanojevic. Version 2, 7 April 2013. Available at: http://www.ers-education.org/guidelines/global-lung-function-initiative/tools/sas-macro.aspx. Accessed 08 December 2015.

# Appendix G: Blood Pressure Normal Levels for Boys and Girls by Age and Height Percentile

## **Blood Pressure Levels for Boys by Age and Height Percentile**

| | ВР | Systolic BP (mmHg) | | | | | | | | Diastolic BP (mmHg) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age<br>(Year) | Percentile | ← Percentile of Height → | | | | | | | | ← Percentile of Height → | | | | | |
| | | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 1 | 50th | 80 | 81 | 83 | 85 | 87 | 88 | 89 | 34 | 35 | 36 | 37 | 38 | 39 | 39 |
| | 90th | 94 | 95 | 97 | 99 | 100 | 102 | 103 | 49 | 50 | 51 | 52 | 53 | 53 | 54 |
| | 95th | 98 | 99 | 101 | 103 | 104 | 106 | 106 | 54 | 54 | 55 | 56 | 57 | 58 | 58 |
| | 99th | 105 | 106 | 108 | 110 | 112 | 113 | 114 | 61 | 62 | 63 | 64 | 65 | 66 | 66 |
| 2 | 50th | 84 | 85 | 87 | 88 | 90 | 92 | 92 | 39 | 40 | 41 | 42 | 43 | 44 | 44 |
| | 90th | 97 | 99 | 100 | 102 | 104 | 105 | 106 | 54 | 55 | 56 | 57 | 58 | 58 | 59 |
| | 95th | 101 | 102 | 104 | 106 | 108 | 109 | 110 | 59 | 59 | 60 | 61 | 62 | 63 | 63 |
| | 99th | 109 | 110 | 111 | 113 | 115 | 117 | 117 | 66 | 67 | 68 | 69 | 70 | 71 | 71 |
| 3 | 50th | 86 | 87 | 89 | 91 | 93 | 94 | 95 | 44 | 44 | 45 | 46 | 47 | 48 | 48 |
| | 90th | 100 | 101 | 103 | 105 | 107 | 108 | 109 | 59 | 59 | 60 | 61 | 62 | 63 | 63 |
| | 95th | 104 | 105 | 107 | 109 | 110 | 112 | 113 | 63 | 63 | 64 | 65 | 66 | 67 | 67 |
| | 99th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 71 | 71 | 72 | 73 | 74 | 75 | 75 |
| 4 | 50th | 88 | 89 | 91 | 93 | 95 | 96 | 97 | 47 | 48 | 49 | 50 | 51 | 51 | 52 |
| | 90th | 102 | 103 | 105 | 107 | 109 | 110 | 111 | 62 | 63 | 64 | 65 | 66 | 66 | 67 |
| | 95th | 106 | 107 | 109 | 111 | 112 | 114 | 115 | 66 | 67 | 68 | 69 | 70 | 71 | 71 |
| | 99th | 113 | 114 | 116 | 118 | 120 | 121 | 122 | 74 | 75 | 76 | 77 | 78 | 78 | 79 |
| 5 | 50th | 90 | 91 | 93 | 95 | 96 | 98 | 98 | 50 | 51 | 52 | 53 | 54 | 55 | 55 |
| | 90th | 104 | 105 | 106 | 108 | 110 | 111 | 112 | 65 | 66 | 67 | 68 | 69 | 69 | 70 |
| | 95th | 108 | 109 | 110 | 112 | 114 | 115 | 116 | 69 | 70 | 71 | 72 | 73 | 74 | 74 |
| | 99th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 77 | 78 | 79 | 80 | 81 | 81 | 82 |
| 6 | 50th | 91 | 92 | 94 | 96 | 98 | 99 | 100 | 53 | 53 | 54 | 55 | 56 | 57 | 57 |
| | 90th | 105 | 106 | 108 | 110 | 111 | 113 | 113 | 68 | 68 | 69 | 70 | 71 | 72 | 72 |
| | 95th | 109 | 110 | 112 | 114 | 115 | 117 | 117 | 72 | 72 | 73 | 74 | 75 | 76 | 76 |
| | 99th | 116 | 117 | 119 | 121 | 123 | 124 | 125 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| 7 | 50th | 92 | 94 | 95 | 97 | 99 | 100 | 101 | 55 | 55 | 56 | 57 | 58 | 59 | 59 |
| | 90th | 106 | 107 | 109 | 111 | 113 | 114 | 115 | 70 | 70 | 71 | 72 | 73 | 74 | 74 |
| | 95th | 110 | 111 | 113 | 115 | 117 | 118 | 119 | 74 | 74 | 75 | 76 | 77 | 78 | 78 |
| | 99th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 82 | 82 | 83 | 84 | 85 | 86 | 86 |
| 8 | 50th | 94 | 95 | 97 | 99 | 100 | 102 | 102 | 56 | 57 | 58 | 59 | 60 | 60 | 61 |
| | 90th | 107 | 109 | 110 | 112 | 114 | 115 | 116 | 71 | 72 | 72 | 73 | 74 | 75 | 76 |
| | 95th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 75 | 76 | 77 | 78 | 79 | 79 | 80 |
| | 99th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 83 | 84 | 85 | 86 | 87 | 87 | 88 |
| 9 | 50th | 95 | 96 | 98 | 100 | 102 | 103 | 104 | 57 | 58 | 59 | 60 | 61 | 61 | 62 |
| | 90th | 109 | 110 | 112 | 114 | 115 | 117 | 118 | 72 | 73 | 74 | 75 | 76 | 76 | 77 |
| | 95th | 113 | 114 | 116 | 118 | 119 | 121 | 121 | 76 | 77 | 78 | 79 | 80 | 81 | 81 |
| | 99th | 120 | 121 | 123 | 125 | 127 | 128 | 129 | 84 | 85 | 86 | 87 | 88 | 88 | 89 |
| 10 | 50th | 97 | 98 | 100 | 102 | 103 | 105 | 106 | 58 | 59 | 60 | 61 | 61 | 62 | 63 |
| | 90th | 111 | 112 | 114 | 115 | 117 | 119 | 119 | 73 | 73 | 74 | 75 | 76 | 77 | 78 |
| | 95th | 115 | 116 | 117 | 119 | 121 | 122 | 123 | 77 | 78 | 79 | 80 | 81 | 81 | 82 |
| | 99th | 122 | 123 | 125 | 127 | 128 | 130 | 130 | 85 | 86 | 86 | 88 | 88 | 89 | 90 |

## Blood Pressure Levels for Boys by Age and Height Percentile (Continued)

| Age<br>(Year) | ВР | Systolic BP (mmHg) | | | | | | | Diastolic BP (mmHg) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Percentile | | ← Percentile of Height → | | | | | | | ← Percentile of Height → | | | | | |
| | $lack \Psi$ | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 11 | 50th | 99 | 100 | 102 | 104 | 105 | 107 | 107 | 59 | 59 | 60 | 61 | 62 | 63 | 63 |
| | 90th | 113 | 114 | 115 | 117 | 119 | 120 | 121 | 74 | 74 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 117 | 118 | 119 | 121 | 123 | 124 | 125 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 124 | 125 | 127 | 129 | 130 | 132 | 132 | 86 | 86 | 87 | 88 | 89 | 90 | 90 |
| 12 | 50th | 101 | 102 | 104 | 106 | 108 | 109 | 110 | 59 | 60 | 61 | 62 | 63 | 63 | 64 |
| | 90th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 74 | 75 | 75 | 76 | 77 | 78 | 79 |
| | 95th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 78 | 79 | 80 | 81 | 82 | 82 | 83 |
| | 99th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 86 | 87 | 88 | 89 | 90 | 90 | 91 |
| 13 | 50th | 104 | 105 | 106 | 108 | 110 | 111 | 112 | 60 | 60 | 61 | 62 | 63 | 64 | 64 |
| | 90th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 75 | 75 | 76 | 77 | 78 | 79 | 79 |
| | 95th | 121 | 122 | 124 | 126 | 128 | 129 | 130 | 79 | 79 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 130 | 131 | 133 | 135 | 136 | 137 | 87 | 87 | 88 | 89 | 90 | 91 | 91 |
| 14 | 50th | 106 | 107 | 109 | 111 | 113 | 114 | 115 | 60 | 61 | 62 | 63 | 64 | 65 | 65 |
| | 90th | 120 | 121 | 123 | 125 | 126 | 128 | 128 | 75 | 76 | 77 | 78 | 79 | 79 | 80 |
| | 95th | 124 | 125 | 127 | 128 | 130 | 132 | 132 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 131 | 132 | 134 | 136 | 138 | 139 | 140 | 87 | 88 | 89 | 90 | 91 | 92 | 92 |
| 15 | 50th | 109 | 110 | 112 | 113 | 115 | 117 | 117 | 61 | 62 | 63 | 64 | 65 | 66 | 66 |
| | 90th | 122 | 124 | 125 | 127 | 129 | 130 | 131 | 76 | 77 | 78 | 79 | 80 | 80 | 81 |
| | 95th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 81 | 81 | 82 | 83 | 84 | 85 | 85 |
| | 99th | 134 | 135 | 136 | 138 | 140 | 142 | 142 | 88 | 89 | 90 | 91 | 92 | 93 | 93 |
| 16 | 50th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 63 | 63 | 64 | 65 | 66 | 67 | 67 |
| | 90th | 125 | 126 | 128 | 130 | 131 | 133 | 134 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 95th | 129 | 130 | 132 | 134 | 135 | 137 | 137 | 82 | 83 | 83 | 84 | 85 | 86 | 87 |
| | 99th | 136 | 137 | 139 | 141 | 143 | 144 | 145 | 90 | 90 | 91 | 92 | 93 | 94 | 94 |
| 17 | 50th | 114 | 115 | 116 | 118 | 120 | 121 | 122 | 65 | 66 | 66 | 67 | 68 | 69 | 70 |
| | 90th | 127 | 128 | 130 | 132 | 134 | 135 | 136 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 95th | 131 | 132 | 134 | 136 | 138 | 139 | 140 | 84 | 85 | 86 | 87 | 87 | 88 | 89 |
| | 99th | 139 | 140 | 141 | 143 | 145 | 146 | 147 | 92 | 93 | 93 | 94 | 95 | 96 | 97 |

BP, blood pressure

For research purposes, the standard deviations in Appendix Table B–1 allow one to compute BP Z-scores and percentiles for boys with height percentiles given in Table 3 (i.e., the 5th,10th, 25th, 50th, 75th, 90th, and 95th percentiles). These height percentiles must be converted to height Z-scores given by (5% = -1.645; 10% = -1.28; 25% = -0.68; 50% = 0; 75% = 0.68; 90% = 1.28%; 95% = 1.645) and then computed according to the methodology in steps 2–4 described in Appendix B. For children with height percentiles other than these, follow steps 1–4 as described in Appendix B.

<sup>\*</sup> The 90th percentile is 1.28 SD, 95th percentile is 1.645 SD, and the 99th percentile is 2.326 SD over the mean.

## **Blood Pressure Levels for Girls by Age and Height Percentile**

| | ВР | Systolic BP (mmHg) | | | | | | | | Diastolic BP (mmHg) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | Percentile | ← Percentile of Height → | | | | | | | | ← Percentile of Height → | | | | | |
| (Year) | | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| I | 50th | 83 | 84 | 85 | 86 | 88 | 89 | 90 | 38 | 39 | 39 | 40 | 41 | 41 | 42 |
| | 90th | 97 | 97 | 98 | 100 | 101 | 102 | 103 | 52 | 53 | 53 | 54 | 55 | 55 | 56 |
| | 95th | 100 | 101 | 102 | 104 | 105 | 106 | 107 | 56 | 57 | 57 | 58 | 59 | 59 | 60 |
| | 99th | 108 | 108 | 109 | 111 | 112 | 113 | 114 | 64 | 64 | 65 | 65 | 66 | 67 | 67 |
| 2 | 50th | 85 | 85 | 87 | 88 | 89 | 91 | 91 | 43 | 44 | 44 | 45 | 46 | 46 | 47 |
| | 90th | 98 | 99 | 100 | 101 | 103 | 104 | 105 | 57 | 58 | 58 | 59 | 60 | 61 | 61 |
| | 95th | 102 | 103 | 104 | 105 | 107 | 108 | 109 | 61 | 62 | 62 | 63 | 64 | 65 | 65 |
| | 99th | 109 | 110 | 111 | 112 | 114 | 115 | 116 | 69 | 69 | 70 | 70 | 71 | 72 | 72 |
| 3 | 50th | 86 | 87 | 88 | 89 | 91 | 92 | 93 | 47 | 48 | 48 | 49 | 50 | 50 | 51 |
| | 90th | 100 | 100 | 102 | 103 | 104 | 106 | 106 | 61 | 62 | 62 | 63 | 64 | 64 | 65 |
| | 95th | 104 | 104 | 105 | 107 | 108 | 109 | 110 | 65 | 66 | 66 | 67 | 68 | 68 | 69 |
| | 99th | 111 | 111 | 113 | 114 | 115 | 116 | 117 | 73 | 73 | 74 | 74 | 75 | 76 | 76 |
| 4 | 50th | 88 | 88 | 90 | 91 | 92 | 94 | 94 | 50 | 50 | 51 | 52 | 52 | 53 | 54 |
| | 90th | 101 | 102 | 103 | 104 | 106 | 107 | 108 | 64 | 64 | 65 | 66 | 67 | 67 | 68 |
| | 95th | 105 | 106 | 107 | 108 | 110 | 111 | 112 | 68 | 68 | 69 | 70 | 71 | 71 | 72 |
| | 99th | 112 | 113 | 114 | 115 | 117 | 118 | 119 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| 5 | 50th | 89 | 90 | 91 | 93 | 94 | 95 | 96 | 52 | 53 | 53 | 54 | 55 | 55 | 56 |
| | 90th | 103 | 103 | 105 | 106 | 107 | 109 | 109 | 66 | 67 | 67 | 68 | 69 | 69 | 70 |
| | 95th | 107 | 107 | 108 | 110 | 111 | 112 | 113 | 70 | 71 | 71 | 72 | 73 | 73 | 74 |
| | 99th | 114 | 114 | 116 | 117 | 118 | 120 | 120 | 78 | 78 | 79 | 79 | 80 | 81 | 81 |
| 6 | 50th | 91 | 92 | 93 | 94 | 96 | 97 | 98 | 54 | 54 | 55 | 56 | 56 | 57 | 58 |
| | 90th | 104 | 105 | 106 | 108 | 109 | 110 | 111 | 68 | 68 | 69 | 70 | 70 | 71 | 72 |
| | 95th | 108 | 109 | 110 | 111 | 113 | 114 | 115 | 72 | 72 | 73 | 74 | 74 | 75 | 76 |
| | 99th | 115 | 116 | 117 | 119 | 120 | 121 | 122 | 80 | 80 | 80 | 81 | 82 | 83 | 83 |
| 7 | 50th | 93 | 93 | 95 | 96 | 97 | 99 | 99 | 55 | 56 | 56 | 57 | 58 | 58 | 59 |
| | 90th | 106 | 107 | 108 | 109 | 111 | 112 | 113 | 69 | 70 | 70 | 71 | 72 | 72 | 73 |
| | 95th | 110 | 111 | 112 | 113 | 115 | 116 | 116 | 73 | 74 | 74 | 75 | 76 | 76 | 77 |
| | 99th | 117 | 118 | 119 | 120 | 122 | 123 | 124 | 81 | 81 | 82 | 82 | 83 | 84 | 84 |
| 8 | 50th | 95 | 95 | 96 | 98 | 99 | 100 | 101 | 57 | 57 | 57 | 58 | 59 | 60 | 60 |
| | 90th | 108 | 109 | 110 | 111 | 113 | 114 | 114 | 71 | 71 | 71 | 72 | 73 | 74 | 74 |
| | 95th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 75 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 99th | 119 | 120 | 121 | 122 | 123 | 125 | 125 | 82 | 82 | 83 | 83 | 84 | 85 | 86 |
| 9 | 50th | 96 | 97 | 98 | 100 | 101 | 102 | 103 | 58 | 58 | 58 | 59 | 60 | 61 | 61 |
| | 90th | 110 | 110 | 112 | 113 | 114 | 116 | 116 | 72 | 72 | 72 | 73 | 74 | 75 | 75 |
| | 95th | 114 | 114 | 115 | 117 | 118 | 119 | 120 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| | 99th | 121 | 121 | 123 | 124 | 125 | 127 | 127 | 83 | 83 | 84 | 84 | 85 | 86 | 87 |
| 10 | 50th | 98 | 99 | 100 | 102 | 103 | 104 | 105 | 59 | 59 | 59 | 60 | 61 | 62 | 62 |
| | 90th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 73 | 73 | 73 | 74 | 75 | 76 | 76 |
| | 95th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 77 | 77 | 77 | 78 | 79 | 80 | 80 |
| | 99th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 84 | 84 | 85 | 86 | 86 | 87 | 88 |

## **Blood Pressure Levels for Girls by Age and Height Percentile (Continued)**

| Age<br>(Year) | ВР | Systolic BP (mmHg) | | | | | | | | Diastolic BP (mmHg) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Percentile | | ← Percentile of Height → | | | | | | | | ← Percentile of Height → | | | | |
| | | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 11 | 50th | 100 | 101 | 102 | 103 | 105 | 106 | 107 | 60 | 60 | 60 | 61 | 62 | 63 | 63 |
| | 90th | 114 | 114 | 116 | 117 | 118 | 119 | 120 | 74 | 74 | 74 | 75 | 76 | 77 | 77 |
| | 95th | 118 | 118 | 119 | 121 | 122 | 123 | 124 | 78 | 78 | 78 | 79 | 80 | 81 | 81 |
| | 99th | 125 | 125 | 126 | 128 | 129 | 130 | 131 | 85 | 85 | 86 | 87 | 87 | 88 | 89 |
| 12 | 50th | 102 | 103 | 104 | 105 | 107 | 108 | 109 | 61 | 61 | 61 | 62 | 63 | 64 | 64 |
| | 90th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 75 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 119 | 120 | 121 | 123 | 124 | 125 | 126 | 79 | 79 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 127 | 127 | 128 | 130 | 131 | 132 | 133 | 86 | 86 | 87 | 88 | 88 | 89 | 90 |
| 13 | 50th | 104 | 105 | 106 | 107 | 109 | 110 | 110 | 62 | 62 | 62 | 63 | 64 | 65 | 65 |
| | 90th | 117 | 118 | 119 | 121 | 122 | 123 | 124 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| | 95th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 80 | 80 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 129 | 130 | 132 | 133 | 134 | 135 | 87 | 87 | 88 | 89 | 89 | 90 | 91 |
| 14 | 50th | 106 | 106 | 107 | 109 | 110 | 111 | 112 | 63 | 63 | 63 | 64 | 65 | 66 | 66 |
| | 90th | 119 | 120 | 121 | 122 | 124 | 125 | 125 | 77 | 77 | 77 | 78 | 79 | 80 | 80 |
| | 95th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 81 | 81 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 130 | 131 | 132 | 133 | 135 | 136 | 136 | 88 | 88 | 89 | 90 | 90 | 91 | 92 |
| 15 | 50th | 107 | 108 | 109 | 110 | 111 | 113 | 113 | 64 | 64 | 64 | 65 | 66 | 67 | 67 |
| | 90th | 120 | 121 | 122 | 123 | 125 | 126 | 127 | 78 | 78 | 78 | 79 | 80 | 81 | 81 |
| | 95th | 124 | 125 | 126 | 127 | 129 | 130 | 131 | 82 | 82 | 82 | 83 | 84 | 85 | 85 |
| | 99th | 131 | 132 | 133 | 134 | 136 | 137 | 138 | 89 | 89 | 90 | 91 | 91 | 92 | 93 |
| 16 | 50th | 108 | 108 | 110 | 111 | 112 | 114 | 114 | 64 | 64 | 65 | 66 | 66 | 67 | 68 |
| | 90th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 78 | 78 | 79 | 80 | 81 | 81 | 82 |
| | 95th | 125 | 126 | 127 | 128 | 130 | 131 | 132 | 82 | 82 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 132 | 133 | 134 | 135 | 137 | 138 | 139 | 90 | 90 | 90 | 91 | 92 | 93 | 93 |
| 17 | 50th | 108 | 109 | 110 | 111 | 113 | 114 | 115 | 64 | 65 | 65 | 66 | 67 | 67 | 68 |
| | 90th | 122 | 122 | 123 | 125 | 126 | 127 | 128 | 78 | 79 | 79 | 80 | 81 | 81 | 82 |
| | 95th | 125 | 126 | 127 | 129 | 130 | 131 | 132 | 82 | 83 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 133 | 133 | 134 | 136 | 137 | 138 | 139 | 90 | 90 | 91 | 91 | 92 | 93 | 93 |

BP, blood pressure

For research purposes, the standard deviations in Appendix Table B-1 allow one to compute BP Z-scores and percentiles for girls with height percentiles given in Table 4 (i.e., the 5th,10th, 25th, 50th, 75th, 90th, and 95th percentiles). These height percentiles must be converted to height Z-scores given by (5% = -1.645; 10% = -1.28; 25% = -0.68; 50% = 0; 75% = 0.68; 90% = 1.28%; 95% = 1.645) and then computed according to the methodology in steps 2-4 described in Appendix B. For children with height percentiles other than these, follow steps 1-4 as described in Appendix B.

<sup>\*</sup> The 90th percentile is 1.28 SD, 95th percentile is 1.645 SD, and the 99th percentile is 2.326 SD over the mean.

# Appendix H: Important Protocol Deviation Programming Rules (Based on the Clinical Database)

The protocol deviations that should be considered as potential IPDs include, but are not limited to:

- Subject entered the study despite violation of an inclusion or exclusion criteria
- Subject received the wrong treatment or incorrect doses
- Subject received excluded concomitant medications
- Subject remained in study despite meeting withdrawal criteria

Occurrence of any of these events should be considered as potential IPDs, but the blinded team should categorize them as IPDs only if they have the potential to affect interpretation of study results. The team should construct rules for identifying IPDs rather than identifying individual subjects with IPDs.

#### Important protocol deviations before first dose

- 1. Inclusion criteria:
  - a. I3: Subjects (males and females) will be between the ages of 2 and 5 years, inclusive, on the date of informed consent (and assent, if applicable) for the relevant study part.
  - b. I4: Subjects who weigh ≥8 kg without shoes and wearing light clothing at the Screening Visit.
  - c. I6: Subjects who are homozygous for *F508del* (genotype to be confirmed at the Screening Visit). If the *CFTR* screening genotype result is not received before Day -1, a previous *CFTR* genotype laboratory report may be used to establish eligibility. Note:
    - Subjects who have been enrolled and whose screening genotype does not confirm study eligibility must be discontinued from the study, as described in Protocol Section 9.5.
    - O This assessment does not need to be repeated for confirmed subjects in Part A who may participate in Part B.

#### 2. Exclusion criteria:

- a. E3: Any of the following abnormal laboratory values at the Screening Visit:
  - o Hemoglobin <10 g/dL
  - o ALT, AST or Total bilirubin >2× ULN
  - o Abnormal renal function defined as glomerular filtration rate ≤45 mL/min/1.73 m² (calculated by the Bedside Schwartz equation)
- b. E5: A standard 12-lead ECG demonstrating QTc >450 msec at the Screening Visit. If QTc exceeds 450 msec at the Screening Visit, the ECG should be repeated 2 more times during the Screening Period, and the average of the 3 QTc values should be used to determine the subject's eligibility.

#### Programming notes:

- o Check if screening QTcF>450 msec at screening, if yes,
- Check whether ECG was repeated 2 more times during the screening period, if no, report as important protocol deviation. If yes,
- o Check whether the average of the 3 QTcF values ≤450msec, if no, report as important protocol deviation.
- c. E6: History of solid organ or hematological transplantation.

#### Important protocol deviations during the treatment period

- 1. Compliance < 80%.
- 2. Prohibited medication not happened during study drug interruption period (prohibited medication treatment period overlaps with study drug treatment period)

#### Programming notes:

- Prohibited medication and study drug should not be taken at the same time/day.
- 3. Nominal Post dose ECGs on Day 1 or Day 15 that are collected before the dosing time on the same visit.

#### Programming note:

- o If the ECG is labeled as post-dose but the actual timing is pre-dose, then it should be reported as important protocol deviation.
- 4. Eye exam is not completed at either Week 24 or the Safety Follow-Up Visit (Week 26).
- 5. Subject received the wrong treatment or incorrect doses.